CLINICAL TRIAL: NCT02328677
Title: ColoCare Transdisciplinary Research in Colorectal Cancer Prognosis
Brief Title: ColoCare Study - Colorectal Cancer Cohort
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: German Cancer Research Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Huntsman Cancer Institute (Other); Cedars-Sinai Medical Center (Other); Washington University School of Medicine (Other); University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 6407; NCT02391597 (obsolete NCT alias)
Record Dates: First submitted 2014-11-17; First posted 2014-12-31 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; rectosigmoid; rectum; colon
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, feces, saliva, FFPE and fresh frozen tissue (multiple sources/locations) from the tumor, DNA, RNA, miRNA, visceral adipose tissue and subcutaneous adipose tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- ColoCare FHCC: Active patient recruitment, follow-up, and multiple specimen collection Repeated sampling at multiple timepoints Longitudinal assessment of biomarkers and health behaviors Recruitment Status August 31, 2023: n=741
- ColoCare Moffitt (affiliated cohort): Active patient recruitment, follow-up, and multiple specimen collection Repeated sampling at multiple timepoints Longitudinal assessment of biomarkers and health behaviors Recruitment Status August 31, 2023: n=1,043
- University Hospital Heidelberg: Active patient recruitment, follow-up, and multiple specimen collection Repeated sampling at multiple timepoints Longitudinal assessment of biomarkers and health behaviors Recruitment Status August 31, 2023: n=773
- ColoCare Huntsman Cancer Institute: Active patient recruitment, follow-up, and multiple specimen collection Repeated sampling at multiple timepoints Longitudinal assessment of biomarkers and health behaviors Recruitment Status August 31, 2023: n=514
- Cedars-Sinai Medical Center: Active patient recruitment, follow-up, and multiple specimen collection Repeated sampling at multiple timepoints Longitudinal assessment of biomarkers and health behaviors Recruitment Status August 31, 2023: n=291
- Washington University School of Medicine in St. Louis: Active patient recruitment, follow-up, and multiple specimen collection Repeated sampling at multiple timepoints Longitudinal assessment of biomarkers and health behaviors Recruitment Status August 31, 2023: n=278
- University of Tennessee: Active patient recruitment, follow-up, and multiple specimen collection Repeated sampling at multiple timepoints Longitudinal assessment of biomarkers and health behaviors Recruitment Status August 31, 2023: n=253

SUMMARY:
ColoCare is an international prospective cohort study of stage I-IV colorectal cancer patients (ICD-10 C18-C20).

DETAILED DESCRIPTION:
The ColoCare Study is a multicenter initiative establishing an international cohort of colorectal cancer (CRC) patients for interdisciplinary studies of CRC prognosis and outcomes with sites at the Fred Hutchinson Cancer Center, Seattle (Washington, USA), H. Lee Moffitt Cancer Center and Research Institute, Tampa (Florida, USA), the University Hospital Heidelberg (Germany), the Huntsman Cancer Institute (Utah, USA), the Cedars-Senai Medical Center (California, USA), University of Washington St. Louis (Missouri, USA), and University of Tennessee (Tennessee, USA).

Aims: The ColoCare Study investigates clinical outcomes, including disease-free and overall survival, predictors of cancer recurrence, survival, health-related quality-of-life and treatment toxicities. In addition, cross-sectional analyses of biomarkers and/or health behaviors are undertaken. Patients will be recruited if their age range is 18-89 years. For patients recruited after 09/01/2021 the age range is between 18-69 years, except if they participate in specific sub-studies or in studies for older cancer patients. Recruitment of patients >70 years was re-initiated after 06/2024 in anticipation of R01 grant funding.

Patients are recruited at baseline (time of first diagnosis) and followed for up to 5 years at regular timepoints (3m, 6m, 12m, 24m, 36m, 48m, 60m). The cohort includes a comprehensive collection of specimens and data. For the U01 renewal phase (start September 2021) we specifically focus on the recruitment of minorities (early-onset patients, African American patients, Hispanic patients) and patients with rectal cancer. Furthermore, we will have an overall focus on questionnaire assessment at baseline, 12, and 60 months and intensive medical chart abstraction 24 months and 60. months after enrollment into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-89 years; for patients recruited after 09/01/2021 the age range is 18-69 years. Recruitment of patients 70 years and older was maintained for specific sub-studies and re-initiated for specific R01 grant funding in ~06/2024
2. Men and women
3. Newly-diagnosed colon or rectal cancer (stages I-IV); CRC in treatment (FHCRC and HCI)
4. English (FHCRC, Moffitt, HCI, Cedars-Sinai, WashU St. Louis) or German (University Hospital Heidelberg)-speaking;
5. mentally/physically able to consent and participate.

Exclusion Criteria:

* if one of the above in not fulfilled
* insufficient language or consent capacity

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ColoCare is an international prospective cohort study of stage I-IV colorectal cancer patients (ICD-10 C18-C20). The ColoCare Consortium is a multicenter initiative of interdisciplinary research on CRC outcome and prognosis, and comprises patient recruitment at 6 sites. Patients are recruited at baseline (time of first diagnosis, time prior to surgery or during treatment (FHCRC and HCI)) and followed for up to 10 years at regular timepoints (3m, 6m, 12m, 24m, 36m, 48m, 60m). The cohort includes a comprehensive collection of biospecimens and data.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-03; Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free and overall survival | up to 10 years
Recurrence | up to 5 years

SECONDARY OUTCOMES:
Health-related quality of life | at 0, 3, 6, 12, 24, 36, 48, 60 months post recruitment
Treatment toxicities | up to 5 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ulrich, MS, PhD, Principal Investigator — Huntsman Cancer Institute; William Grady, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Christopher Li, MD, Principal Investigator — Fred Hutchinson Cancer Center; Doratha Byrd, PhD, Principal Investigator — Lee H. Moffitt Cancer Center; Jane Figueiredo, PhD, Principal Investigator — Cedars-Sinai Medical Center; David Shibata, MD, Principal Investigator — University of Tennesee; Adetunji T. Toriola, MD, PhD, Principal Investigator — Washington University School of Medicine; Biljana Gigic, PhD, Principal Investigator — Heidelberg University
Locations (7):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Lee H. Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - University of Tennessee, Knoxville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - FHCRC, Seattle, Washington
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Himbert C, Delphan M, Scherer D, Bowers LW, Hursting S, Ulrich CM. Signals from the Adipose Microenvironment and the Obesity-Cancer Link-A Systematic Review. Cancer Prev Res (Phila). 2017 Sep;10(9):494-506. doi: 10.1158/1940-6207.CAPR-16-0322. PMID 28864539
- [Background] Ulrich CM, Himbert C, Holowatyj AN, Hursting SD. Energy balance and gastrointestinal cancer: risk, interventions, outcomes and mechanisms. Nat Rev Gastroenterol Hepatol. 2018 Nov;15(11):683-698. doi: 10.1038/s41575-018-0053-2. PMID 30158569
- [Background] Zhang P, Holowatyj AN, Roy T, Pronovost SM, Marchetti M, Liu H, Ulrich CM, Edgar BA. An SH3PX1-Dependent Endocytosis-Autophagy Network Restrains Intestinal Stem Cell Proliferation by Counteracting EGFR-ERK Signaling. Dev Cell. 2019 May 20;49(4):574-589.e5. doi: 10.1016/j.devcel.2019.03.029. Epub 2019 Apr 18. PMID 31006650
- [Background] Yu B, Zanetti KA, Temprosa M, Albanes D, Appel N, Barrera CB, Ben-Shlomo Y, Boerwinkle E, Casas JP, Clish C, Dale C, Dehghan A, Derkach A, Eliassen AH, Elliott P, Fahy E, Gieger C, Gunter MJ, Harada S, Harris T, Herr DR, Herrington D, Hirschhorn JN, Hoover E, Hsing AW, Johansson M, Kelly RS, Khoo CM, Kivimaki M, Kristal BS, Langenberg C, Lasky-Su J, Lawlor DA, Lotta LA, Mangino M, Le Marchand L, Mathe E, Matthews CE, Menni C, Mucci LA, Murphy R, Oresic M, Orwoll E, Ose J, Pereira AC, Playdon MC, Poston L, Price J, Qi Q, Rexrode K, Risch A, Sampson J, Seow WJ, Sesso HD, Shah SH, Shu XO, Smith GCS, Sovio U, Stevens VL, Stolzenberg-Solomon R, Takebayashi T, Tillin T, Travis R, Tzoulaki I, Ulrich CM, Vasan RS, Verma M, Wang Y, Wareham NJ, Wong A, Younes N, Zhao H, Zheng W, Moore SC. The Consortium of Metabolomics Studies (COMETS): Metabolomics in 47 Prospective Cohort Studies. Am J Epidemiol. 2019 Jun 1;188(6):991-1012. doi: 10.1093/aje/kwz028. PMID 31155658
- [Background] Playdon MC, Joshi AD, Tabung FK, Cheng S, Henglin M, Kim A, Lin T, van Roekel EH, Huang J, Krumsiek J, Wang Y, Mathe E, Temprosa M, Moore S, Chawes B, Eliassen AH, Gsur A, Gunter MJ, Harada S, Langenberg C, Oresic M, Perng W, Seow WJ, Zeleznik OA. Metabolomics Analytics Workflow for Epidemiological Research: Perspectives from the Consortium of Metabolomics Studies (COMETS). Metabolites. 2019 Jul 17;9(7):145. doi: 10.3390/metabo9070145. PMID 31319517
- [Background] Holowatyj AN, Lewis MA, Pannier ST, Kirchhoff AC, Hardikar S, Figueiredo JC, Huang LC, Shibata D, Schmit SL, Ulrich CM. Clinicopathologic and Racial/Ethnic Differences of Colorectal Cancer Among Adolescents and Young Adults. Clin Transl Gastroenterol. 2019 Jul;10(7):e00059. doi: 10.14309/ctg.0000000000000059. PMID 31259751
- [Background] Zhang P, Holowatyj AN, Ulrich CM, Edgar BA. Tumor suppressive autophagy in intestinal stem cells controls gut homeostasis. Autophagy. 2019 Sep;15(9):1668-1670. doi: 10.1080/15548627.2019.1633863. Epub 2019 Jun 20. PMID 31213134
- [Result] Simon LH, Saviers-Steiger C, Dunston ER, Galyean P, Kimball ER, Mendez J, Zickmund SL, Hansen PA, Ulrich CM, LaStayo PC, Steinberg D, Noren CS, Finch A, Seckinger L, Braun E, Chipman J, Brownson KE, Oza S, Coletta AM. Feasibility and acceptability of the Comprehensive Oncology Rehabilitation and Exercise (CORE) clinical workflow algorithm in patients with newly diagnosed stage I-III breast cancer who undergo surgery as first-line treatment. Cancer. 2025 May 1;131(9):e35798. doi: 10.1002/cncr.35798. PMID 40289623
- [Result] Ulrich CM, Himbert C, Barnes CA, Boucher KM, Daniels B, Bandera VM, Ligibel JA, Wetter DW, Hess R, Kim J, Lundberg K, Mitzman B, Marcus R, Finlayson SRG, LaStayo PC, Varghese TK Jr. Precision Exercise Effect on Fatigue and Function in Lung Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 May 1;160(5):495-519. doi: 10.1001/jamasurg.2025.0130. PMID 40072448
- [Result] Saez-Clarke E, Otto AK, Prinsloo S, Natori A, Wagner RW, Gomez TI, Ochoa JM, Tworoger SS, Ulrich CM, Hathaway CA, Peoples AR, Antoni MH, Bower JE, Cohen L, Penedo FJ. Development and initial psychometric evaluation of a COVID-related psychosocial experiences questionnaire for cancer survivors. Qual Life Res. 2023 Dec;32(12):3475-3494. doi: 10.1007/s11136-023-03456-4. Epub 2023 Jun 26. PMID 37358738
- [Result] Watts EL, Gonzales TI, Strain T, Saint-Maurice PF, Bishop DT, Chanock SJ, Johansson M, Keku TO, Le Marchand L, Moreno V, Newcomb PA, Newton CC, Pai RK, Purdue MP, Ulrich CM, Smith-Byrne K, Van Guelpen B; PRACTICAL consortium, CRUK, BPC3, CAPS, PEGASUS; Day FR, Wijndaele K, Wareham NJ, Matthews CE, Moore SC, Brage S. Observational and genetic associations between cardiorespiratory fitness and cancer: a UK Biobank and international consortia study. Br J Cancer. 2024 Jan;130(1):114-124. doi: 10.1038/s41416-023-02489-3. Epub 2023 Dec 6. PMID 38057395
- [Result] Siegel EM, Ulrich CM, Shibata D. Risk Stratification for Early-onset Colorectal Cancer Screening: Are We Ready for Implementation? Cancer Prev Res (Phila). 2023 Sep 1;16(9):479-481. doi: 10.1158/1940-6207.CAPR-23-0239. PMID 37655450
- [Result] Hiensch AE, Beckhaus J, Witlox L, Monninkhof EM, Schagen SB, van Vulpen JK, Sweegers MG, Newton RU, Aaronson NK, Galvao DA, Steindorf K, Stuiver MM, Mesters I, Knoop H, Goedendorp MM, Bohus M, Thorsen L, Schulz KH, Schmidt ME, Ulrich CM, Sonke GS, van Harten WH, Winters-Stone KM, Velthuis MJ, Taaffe DR, van Mechelen W, Kersten MJ, Nollet F, Wiskemann J, Buffart LM, May AM. Moderators of exercise effects on self-reported cognitive functioning in cancer survivors: an individual participant data meta-analysis. J Cancer Surviv. 2024 Oct;18(5):1492-1503. doi: 10.1007/s11764-023-01392-3. Epub 2023 May 9. PMID 37160571
- [Result] Jin N, Hoyd R, Yilmaz AS, Zhu J, Liu Y, Singh MJ, Grencewicz D, Mo X, Kalady M, Rosenberg D, Dravillas CE, Singer EA, Carpten JD, Chan CH, Churchman ML, Denko NC, Di Clemente F, Dodd RD, Eljilany I, Fei N, Hardikar S, Ikeguchi AP, Ma A, Ma Q, McCarter MD, Osman AE, Riedlinger G, Robinson LA, Schneider BP, Tarhini AA, Tinoco G, Figueiredo J, Zakharia Y, Ulrich CM, Tan AC, Spakowicz D. Epigenetic Modulation, Intra-tumoral Microbiome and Immunity in Early Onset Colorectal Cancer. bioRxiv [Preprint]. 2025 Apr 2:2025.03.28.645992. doi: 10.1101/2025.03.28.645992. PMID 40236026
- [Result] Holthuijsen DDB, Rijnhart JJM, Bours MJL, van Roekel EH, Ueland PM, Breukink SO, Janssen-Heijnen MLG, Konsten JL, Keulen ETP, McCann A, Brezina S, Gigic B, Ulrich CM, Weijenberg MP, Eussen SJPM. Longitudinal associations of dietary intake with fatigue in colorectal cancer survivors up to 1 year post-treatment, and the potential mediating role of the kynurenine pathway. Brain Behav Immun. 2025 May;126:144-159. doi: 10.1016/j.bbi.2025.02.003. Epub 2025 Feb 7. PMID 39922470
- [Result] Holthuijsen DDB, van Roekel EH, Bours MJL, Ueland PM, Breukink SO, Janssen-Heijnen MLG, Konsten JL, Keulen ETP, McCann A, Brezina S, Gigic B, Kok DE, Ulrich CM, Weijenberg MP, Eussen SJPM. Modeling how iso-caloric macronutrient substitutions are longitudinally associated with plasma kynurenines in colorectal cancer survivors up to 12 months post-treatment. J Nutr Biochem. 2025 Jul;141:109910. doi: 10.1016/j.jnutbio.2025.109910. Epub 2025 Mar 28. PMID 40158742
- [Result] Viskochil RH, Lin T, Gigic B, Himbert C, Bandera VM, Skender S, Holowatyj AN, Schrotz-King P, Steindorf K, Strehli I, Mutch MG, Chao D, Toriola AT, Shibata D, Siegel EM, Li CI, Hardikar S, Peoples AR, Figueiredo JC, Schneider M, Ulrich CM, Ose J. Sedentary behavior and physical activity one year after colorectal cancer diagnosis: results from the ColoCare Study. J Cancer Surviv. 2025 Feb 22. doi: 10.1007/s11764-025-01756-x. Online ahead of print. PMID 39985691
- [Result] Alduhayh S, Laskar RS, Jiang X, Zhu Z, Vincent EE, Constantinescu AE, Buchanan DD, Grant RC, Phipps AI, Brenner H, Huang WY, Kweon SS, Li L, Pearlman R, Castellvi-Bel S, Gruber SB, Li CI, Pellatt A, Platz EA, Van Guelpen B, Zheng W, Chan AT, Figueiredo JC, Ogino S, Ulrich CM, Gunter MJ, Haycock P, Severi G, Murphy N, Dimou N. Association of Genetic Liability to Allergic Diseases with Overall and Early-Onset Colorectal Cancer Risk: A Mendelian Randomization Study. Cancer Epidemiol Biomarkers Prev. 2025 May 2;34(5):722-736. doi: 10.1158/1055-9965.EPI-24-0970. PMID 39982694
- [Result] Byrd DA, Damerell V, Gomez Morales MF, Hogue SR, Lin T, Ose J, Himbert C, Ilozumba MN, Kahlert C, Shibata D, Toriola AT, Li CI, Figueiredo J, Stephens WZ, Warby CA, Hardikar S, Siegel EM, Round J, Ulrich CM, Gigic B. The gut microbiome is associated with disease-free survival in stage I-III colorectal cancer patients. Int J Cancer. 2025 Jul 1;157(1):64-73. doi: 10.1002/ijc.35342. Epub 2025 Jan 31. PMID 39887373
- [Result] Ilozumba MN, Lin T, Hardikar S, Byrd DA, Round JL, Stephens WZ, Holowatyj AN, Warby CA, Damerell V, Li CI, Figueiredo JC, Toriola AT, Shibata D, Fillmore GC, Pickron B, Siegel EM, Kahlert C, Florou V, Gigic B, Ose J, Ulrich CM. Fusobacterium nucleatum Abundance is Associated with Cachexia in Colorectal Cancer Patients: The ColoCare Study. Cancer Med. 2024 Nov;13(22):e70431. doi: 10.1002/cam4.70431. PMID 39587707
- [Result] Noriega Esquives BS, Natori A, Antoni MH, Otto AK, Prinsloo S, Wagner RW, Gomez TI, Hathaway CA, Ulrich CM, Peoples AR, Cohen L, Penedo FJ. The impact of negative COVID-19 experiences on cancer survivors' health-related quality of life and psychological distress: a moderated mediation model. Front Psychol. 2024 Sep 12;15:1423106. doi: 10.3389/fpsyg.2024.1423106. eCollection 2024. PMID 39351113
- [Result] O'Neil B, Dindinger-Hill K, Gill H, Coombs L, Haaland B, Ying J, Nelson RE, McPherson J, Kirchhoff AC, Ulrich CM, Huber J, Beck A, Mooney K. Cost and Utilization Outcomes in Huntsman at Home, a Novel Oncology Hospital at Home Program. J Am Med Dir Assoc. 2024 Apr;25(4):610-613. doi: 10.1016/j.jamda.2023.06.030. Epub 2023 Aug 1. PMID 37541650
- [Result] Gauderman WJ, Fu Y, Queme B, Kawaguchi E, Wang Y, Morrison J, Brenner H, Chan A, Gruber SB, Keku T, Li L, Moreno V, Pellatt AJ, Peters U, Samadder NJ, Schmit SL, Ulrich CM, Um C, Wu A, Lewinger JP, Drew DA, Mi H. Pathway Polygenic Risk Scores (pPRS) for the Analysis of Gene-environment Interaction. bioRxiv [Preprint]. 2024 Dec 19:2024.12.16.628610. doi: 10.1101/2024.12.16.628610. PMID 39763728
- [Result] Ose DJ, Adediran E, Mark B, Ocier K, Dunson WA Jr, Turner C, Taylor B, Svoboda K, Post AR, Leiser J, Colman H, Ulrich CM, Hashibe M. The association of diabetes mellitus and routinely collected patient-reported outcomes in patients with cancer. A real-world cohort study. Cancer Med. 2024 Oct;13(20):e70246. doi: 10.1002/cam4.70246. PMID 39445809
- [Result] Damerell V, Klaassen-Dekker N, Brezina S, Ose J, Ulvik A, van Roekel EH, Holowatyj AN, Baierl A, Bohm J, Bours MJL, Brenner H, de Wilt JHW, Grady WM, Habermann N, Hoffmeister M, Keski-Rahkonen P, Lin T, Schirmacher P, Schrotz-King P, Ulrich AB, van Duijnhoven FJB, Warby CA, Shibata D, Toriola AT, Figueiredo JC, Siegel EM, Li CI, Gsur A, Kampman E, Schneider M, Ueland PM, Weijenberg MP, Ulrich CM, Kok DE, Gigic B; FOCUS Consortium. Circulating tryptophan-kynurenine pathway metabolites are associated with all-cause mortality among patients with stage I-III colorectal cancer. Int J Cancer. 2025 Feb 1;156(3):552-565. doi: 10.1002/ijc.35183. Epub 2024 Sep 23. PMID 39308420
- [Result] Hattangady NG, Carter K, Maroni-Rana B, Wang T, Ayers JL, Yu M, Grady WM. Mapping the core senescence phenotype of primary human colon fibroblasts. Aging (Albany NY). 2024 Feb 21;16(4):3068-3087. doi: 10.18632/aging.205577. Epub 2024 Feb 21. PMID 38385965
- [Result] Clark W, Siegel EM, Chen YA, Zhao X, Parsons CM, Hernandez JM, Weber J, Thareja S, Choi J, Shibata D. Quantitative measures of visceral adiposity and body mass index in predicting rectal cancer outcomes after neoadjuvant chemoradiation. J Am Coll Surg. 2013 Jun;216(6):1070-81. doi: 10.1016/j.jamcollsurg.2013.01.007. Epub 2013 Mar 21. PMID 23523147
- [Result] Ulrich CM, Toriola AT, Siegel EM, Brenner H, Chang-Claude J, Abbenhardt C, Kotzmann J, Song X, Owen RW, Hoffmeister M, Becher H, Shibata D, Vickers K, Rush SK, Makar K, Wurtele G, Haubner R, Sellers TA, Grady W. Plasma 25-hydroxyvitamin D3, folate and vitamin B12 biomarkers among international colorectal cancer patients: a pilot study. J Nutr Sci. 2013 Apr 9;2:e9. doi: 10.1017/jns.2012.28. eCollection 2013. PMID 25191595
- [Result] Sherwood AM, Emerson RO, Scherer D, Habermann N, Buck K, Staffa J, Desmarais C, Halama N, Jaeger D, Schirmacher P, Herpel E, Kloor M, Ulrich A, Schneider M, Ulrich CM, Robins H. Tumor-infiltrating lymphocytes in colorectal tumors display a diversity of T cell receptor sequences that differ from the T cells in adjacent mucosal tissue. Cancer Immunol Immunother. 2013 Sep;62(9):1453-61. doi: 10.1007/s00262-013-1446-2. Epub 2013 Jun 16. PMID 23771160
- [Result] Luo Y, Wong CJ, Kaz AM, Dzieciatkowski S, Carter KT, Morris SM, Wang J, Willis JE, Makar KW, Ulrich CM, Lutterbaugh JD, Shrubsole MJ, Zheng W, Markowitz SD, Grady WM. Differences in DNA methylation signatures reveal multiple pathways of progression from adenoma to colorectal cancer. Gastroenterology. 2014 Aug;147(2):418-29.e8. doi: 10.1053/j.gastro.2014.04.039. Epub 2014 Apr 30. PMID 24793120
- [Result] Zeller G, Tap J, Voigt AY, Sunagawa S, Kultima JR, Costea PI, Amiot A, Bohm J, Brunetti F, Habermann N, Hercog R, Koch M, Luciani A, Mende DR, Schneider MA, Schrotz-King P, Tournigand C, Tran Van Nhieu J, Yamada T, Zimmermann J, Benes V, Kloor M, Ulrich CM, von Knebel Doeberitz M, Sobhani I, Bork P. Potential of fecal microbiota for early-stage detection of colorectal cancer. Mol Syst Biol. 2014 Nov 28;10(11):766. doi: 10.15252/msb.20145645. PMID 25432777
- [Result] Ristau J, Staffa J, Schrotz-King P, Gigic B, Makar KW, Hoffmeister M, Brenner H, Ulrich A, Schneider M, Ulrich CM, Habermann N. Suitability of circulating miRNAs as potential prognostic markers in colorectal cancer. Cancer Epidemiol Biomarkers Prev. 2014 Dec;23(12):2632-7. doi: 10.1158/1055-9965.EPI-14-0556. PMID 25472670
- [Result] Skender S, Schrotz-King P, Bohm J, Abbenhardt C, Gigic B, Chang-Claude J, Siegel EM, Steindorf K, Ulrich CM. Repeat physical activity measurement by accelerometry among colorectal cancer patients--feasibility and minimal number of days of monitoring. BMC Res Notes. 2015 Jun 6;8:222. doi: 10.1186/s13104-015-1168-y. PMID 26048683
- [Result] Liesenfeld DB, Grapov D, Fahrmann JF, Salou M, Scherer D, Toth R, Habermann N, Bohm J, Schrotz-King P, Gigic B, Schneider M, Ulrich A, Herpel E, Schirmacher P, Fiehn O, Lampe JW, Ulrich CM. Metabolomics and transcriptomics identify pathway differences between visceral and subcutaneous adipose tissue in colorectal cancer patients: the ColoCare study. Am J Clin Nutr. 2015 Aug;102(2):433-43. doi: 10.3945/ajcn.114.103804. Epub 2015 Jul 8. PMID 26156741
- [Result] Garcia-Albeniz X, Rudolph A, Hutter C, White E, Lin Y, Rosse SA, Figueiredo JC, Harrison TA, Jiao S, Brenner H, Casey G, Hudson TJ, Thornquist M, Le Marchand L, Potter J, Slattery ML, Zanke B, Baron JA, Caan BJ, Chanock SJ, Berndt SI, Stelling D, Fuchs CS, Hoffmeister M, Butterbach K, Du M, James Gauderman W, Gunter MJ, Lemire M, Ogino S, Lin J, Hayes RB, Haile RW, Schoen RE, Warnick GS, Jenkins MA, Thibodeau SN, Schumacher FR, Lindor NM, Kolonel LN, Hopper JL, Gong J, Seminara D, Pflugeisen BM, Ulrich CM, Qu C, Duggan D, Cotterchio M, Campbell PT, Carlson CS, Newcomb PA, Giovannucci E, Hsu L, Chan AT, Peters U, Chang-Claude J. CYP24A1 variant modifies the association between use of oestrogen plus progestogen therapy and colorectal cancer risk. Br J Cancer. 2016 Jan 19;114(2):221-9. doi: 10.1038/bjc.2015.443. Epub 2016 Jan 14. PMID 26766742
- [Result] Skender S, Ose J, Chang-Claude J, Paskow M, Bruhmann B, Siegel EM, Steindorf K, Ulrich CM. Accelerometry and physical activity questionnaires - a systematic review. BMC Public Health. 2016 Jun 16;16:515. doi: 10.1186/s12889-016-3172-0. PMID 27306667
- [Result] Bohm J, Pianka F, Stuttgen N, Rho J, Gigic B, Zhang Y, Habermann N, Schrotz-King P, Abbenhardt-Martin C, Zielske L, Lampe PD, Ulrich A, Diener MK, Ulrich CM. Discovery of novel plasma proteins as biomarkers for the development of incisional hernias after midline incision in patients with colorectal cancer: The ColoCare study. Surgery. 2017 Mar;161(3):808-817. doi: 10.1016/j.surg.2016.08.025. Epub 2016 Oct 13. PMID 27745870
- [Result] Gong J, Hutter CM, Newcomb PA, Ulrich CM, Bien SA, Campbell PT, Baron JA, Berndt SI, Bezieau S, Brenner H, Casey G, Chan AT, Chang-Claude J, Du M, Duggan D, Figueiredo JC, Gallinger S, Giovannucci EL, Haile RW, Harrison TA, Hayes RB, Hoffmeister M, Hopper JL, Hudson TJ, Jeon J, Jenkins MA, Kocarnik J, Kury S, Le Marchand L, Lin Y, Lindor NM, Nishihara R, Ogino S, Potter JD, Rudolph A, Schoen RE, Schrotz-King P, Seminara D, Slattery ML, Thibodeau SN, Thornquist M, Toth R, Wallace R, White E, Jiao S, Lemire M, Hsu L, Peters U; CCFR and GECCO. Genome-Wide Interaction Analyses between Genetic Variants and Alcohol Consumption and Smoking for Risk of Colorectal Cancer. PLoS Genet. 2016 Oct 10;12(10):e1006296. doi: 10.1371/journal.pgen.1006296. eCollection 2016 Oct. PMID 27723779
- [Result] Nattenmueller J, Hoegenauer H, Boehm J, Scherer D, Paskow M, Gigic B, Schrotz-King P, Grenacher L, Ulrich C, Kauczor HU. CT-based compartmental quantification of adipose tissue versus body metrics in colorectal cancer patients. Eur Radiol. 2016 Nov;26(11):4131-4140. doi: 10.1007/s00330-016-4231-8. Epub 2016 Feb 6. PMID 26852215
- [Result] Skender S, Bohm J, Schrotz-King P, Chang-Claude J, Siegel EM, Steindorf K, Owen RW, Ose J, Hoffmeister M, Brenner H, Ulrich CM. Plasma 25-Hydroxyvitamin D3 Levels in Colorectal Cancer Patients and Associations with Physical Activity. Nutr Cancer. 2017 Feb-Mar;69(2):229-237. doi: 10.1080/01635581.2017.1265131. Epub 2017 Jan 17. PMID 28094599
- [Result] Ozoya OO, Siegel EM, Srikumar T, Bloomer AM, DeRenzis A, Shibata D. Quantitative Assessment of Visceral Obesity and Postoperative Colon Cancer Outcomes. J Gastrointest Surg. 2017 Mar;21(3):534-542. doi: 10.1007/s11605-017-3362-9. Epub 2017 Jan 18. PMID 28101721
- [Result] Ulrich CM, Gigic B, Bohm J, Ose J, Viskochil R, Schneider M, Colditz GA, Figueiredo JC, Grady WM, Li CI, Shibata D, Siegel EM, Toriola AT, Ulrich A. The ColoCare Study: A Paradigm of Transdisciplinary Science in Colorectal Cancer Outcomes. Cancer Epidemiol Biomarkers Prev. 2019 Mar;28(3):591-601. doi: 10.1158/1055-9965.EPI-18-0773. Epub 2018 Dec 6. PMID 30523039
- [Result] Yuan Z, Baker K, Redman MW, Wang L, Adams SV, Yu M, Dickinson B, Makar K, Ulrich N, Bohm J, Wurscher M, Westerhoff M, Medwell S, Moonka R, Sinanan M, Fichera A, Vickers K, Grady WM. Dynamic plasma microRNAs are biomarkers for prognosis and early detection of recurrence in colorectal cancer. Br J Cancer. 2017 Oct 10;117(8):1202-1210. doi: 10.1038/bjc.2017.266. Epub 2017 Aug 15. PMID 28809863
- [Result] Barrow TM, Klett H, Toth R, Bohm J, Gigic B, Habermann N, Scherer D, Schrotz-King P, Skender S, Abbenhardt-Martin C, Zielske L, Schneider M, Ulrich A, Schirmacher P, Herpel E, Brenner H, Busch H, Boerries M, Ulrich CM, Michels KB. Smoking is associated with hypermethylation of the APC 1A promoter in colorectal cancer: the ColoCare Study. J Pathol. 2017 Nov;243(3):366-375. doi: 10.1002/path.4955. Epub 2017 Sep 29. PMID 28791728
- [Result] Gigic B, Boeing H, Toth R, Bohm J, Habermann N, Scherer D, Schrotz-King P, Abbenhardt-Martin C, Skender S, Brenner H, Chang-Claude J, Hoffmeister M, Syrjala K, Jacobsen PB, Schneider M, Ulrich A, Ulrich CM. Associations Between Dietary Patterns and Longitudinal Quality of Life Changes in Colorectal Cancer Patients: The ColoCare Study. Nutr Cancer. 2018 Jan;70(1):51-60. doi: 10.1080/01635581.2018.1397707. Epub 2017 Dec 15. PMID 29244538
- [Result] Delphan M, Lin T, Liesenfeld DB, Nattenmuller J, Bohm JT, Gigic B, Habermann N, Zielske L, Schrotz-King P, Schneider M, Ulrich A, Kauczor HU, Ulrich CM, Ose J. Associations of branched-chain amino acids with parameters of energy balance and survival in colorectal cancer patients: Results from the ColoCare Study. Metabolomics. 2018 Mar;2018(14):22. doi: 10.1007/s11306-017-1314-8. Epub 2018 Jan 31. PMID 29706852
- [Result] Babaei M, Jansen L, Balavarca Y, Sjovall A, Bos A, van de Velde T, Moreau M, Liberale G, Goncalves AF, Bento MJ, Ulrich CM, Schrotz-King P, Lemmens V, Glimelius B, Brenner H. Neoadjuvant Therapy in Rectal Cancer Patients With Clinical Stage II to III Across European Countries: Variations and Outcomes. Clin Colorectal Cancer. 2018 Mar;17(1):e129-e142. doi: 10.1016/j.clcc.2017.09.002. Epub 2017 Sep 28. PMID 29074354
- [Result] Babaei M, Balavarca Y, Jansen L, Lemmens V, van Erning FN, van Eycken L, Vaes E, Sjovall A, Glimelius B, Ulrich CM, Schrotz-King P, Brenner H. Administration of adjuvant chemotherapy for stage II-III colon cancer patients: An European population-based study. Int J Cancer. 2018 Apr 1;142(7):1480-1489. doi: 10.1002/ijc.31168. Epub 2017 Dec 4. PMID 29159866
- [Result] Paleari L, Burhenne J, Weiss J, Foersch S, Roth W, Parodi A, Gnant M, Bachleitner-Hofmann T, Scherer D, Ulrich CM, Stabuc B, Puntoni M, Coccia G, Petrera M, Haefeli WE, DeCensi A. High Accumulation of Metformin in Colonic Tissue of Subjects With Diabetes or the Metabolic Syndrome. Gastroenterology. 2018 Apr;154(5):1543-1545. doi: 10.1053/j.gastro.2017.12.040. Epub 2018 Mar 8. No abstract available. PMID 29526732
- [Result] Hu C , Shi Y , Sun C , Liang S , Bao S , Pang M . Facile preparation of ion-doped poly(p-phenylenediamine) nanoparticles for photothermal therapy. Chem Commun (Camb). 2018 May 8;54(38):4862-4865. doi: 10.1039/c8cc01100a. PMID 29697104
- [Result] Schmit SL, Edlund CK, Schumacher FR, Gong J, Harrison TA, Huyghe JR, Qu C, Melas M, Van Den Berg DJ, Wang H, Tring S, Plummer SJ, Albanes D, Alonso MH, Amos CI, Anton K, Aragaki AK, Arndt V, Barry EL, Berndt SI, Bezieau S, Bien S, Bloomer A, Boehm J, Boutron-Ruault MC, Brenner H, Brezina S, Buchanan DD, Butterbach K, Caan BJ, Campbell PT, Carlson CS, Castelao JE, Chan AT, Chang-Claude J, Chanock SJ, Cheng I, Cheng YW, Chin LS, Church JM, Church T, Coetzee GA, Cotterchio M, Cruz Correa M, Curtis KR, Duggan D, Easton DF, English D, Feskens EJM, Fischer R, FitzGerald LM, Fortini BK, Fritsche LG, Fuchs CS, Gago-Dominguez M, Gala M, Gallinger SJ, Gauderman WJ, Giles GG, Giovannucci EL, Gogarten SM, Gonzalez-Villalpando C, Gonzalez-Villalpando EM, Grady WM, Greenson JK, Gsur A, Gunter M, Haiman CA, Hampe J, Harlid S, Harju JF, Hayes RB, Hofer P, Hoffmeister M, Hopper JL, Huang SC, Huerta JM, Hudson TJ, Hunter DJ, Idos GE, Iwasaki M, Jackson RD, Jacobs EJ, Jee SH, Jenkins MA, Jia WH, Jiao S, Joshi AD, Kolonel LN, Kono S, Kooperberg C, Krogh V, Kuehn T, Kury S, LaCroix A, Laurie CA, Lejbkowicz F, Lemire M, Lenz HJ, Levine D, Li CI, Li L, Lieb W, Lin Y, Lindor NM, Liu YR, Loupakis F, Lu Y, Luh F, Ma J, Mancao C, Manion FJ, Markowitz SD, Martin V, Matsuda K, Matsuo K, McDonnell KJ, McNeil CE, Milne R, Molina AJ, Mukherjee B, Murphy N, Newcomb PA, Offit K, Omichessan H, Palli D, Cotore JPP, Perez-Mayoral J, Pharoah PD, Potter JD, Qu C, Raskin L, Rennert G, Rennert HS, Riggs BM, Schafmayer C, Schoen RE, Sellers TA, Seminara D, Severi G, Shi W, Shibata D, Shu XO, Siegel EM, Slattery ML, Southey M, Stadler ZK, Stern MC, Stintzing S, Taverna D, Thibodeau SN, Thomas DC, Trichopoulou A, Tsugane S, Ulrich CM, van Duijnhoven FJB, van Guelpan B, Vijai J, Virtamo J, Weinstein SJ, White E, Win AK, Wolk A, Woods M, Wu AH, Wu K, Xiang YB, Yen Y, Zanke BW, Zeng YX, Zhang B, Zubair N, Kweon SS, Figueiredo JC, Zheng W, Marchand LL, Lindblom A, Moreno V, Peters U, Casey G, Hsu L, Conti DV, Gruber SB. Novel Common Genetic Susceptibility Loci for Colorectal Cancer. J Natl Cancer Inst. 2019 Feb 1;111(2):146-157. doi: 10.1093/jnci/djy099. PMID 29917119
- [Result] Rosenthal EA, Shirts BH, Amendola LM, Horike-Pyne M, Robertson PD, Hisama FM, Bennett RL, Dorschner MO, Nickerson DA, Stanaway IB, Nassir R, Vickers KT, Li C, Grady WM, Peters U, Jarvik GP; NHLBI GO Exome Sequencing Project. Rare loss of function variants in candidate genes and risk of colorectal cancer. Hum Genet. 2018 Oct;137(10):795-806. doi: 10.1007/s00439-018-1938-4. Epub 2018 Sep 28. PMID 30267214
- [Result] Huyghe JR, Bien SA, Harrison TA, Kang HM, Chen S, Schmit SL, Conti DV, Qu C, Jeon J, Edlund CK, Greenside P, Wainberg M, Schumacher FR, Smith JD, Levine DM, Nelson SC, Sinnott-Armstrong NA, Albanes D, Alonso MH, Anderson K, Arnau-Collell C, Arndt V, Bamia C, Banbury BL, Baron JA, Berndt SI, Bezieau S, Bishop DT, Boehm J, Boeing H, Brenner H, Brezina S, Buch S, Buchanan DD, Burnett-Hartman A, Butterbach K, Caan BJ, Campbell PT, Carlson CS, Castellvi-Bel S, Chan AT, Chang-Claude J, Chanock SJ, Chirlaque MD, Cho SH, Connolly CM, Cross AJ, Cuk K, Curtis KR, de la Chapelle A, Doheny KF, Duggan D, Easton DF, Elias SG, Elliott F, English DR, Feskens EJM, Figueiredo JC, Fischer R, FitzGerald LM, Forman D, Gala M, Gallinger S, Gauderman WJ, Giles GG, Gillanders E, Gong J, Goodman PJ, Grady WM, Grove JS, Gsur A, Gunter MJ, Haile RW, Hampe J, Hampel H, Harlid S, Hayes RB, Hofer P, Hoffmeister M, Hopper JL, Hsu WL, Huang WY, Hudson TJ, Hunter DJ, Ibanez-Sanz G, Idos GE, Ingersoll R, Jackson RD, Jacobs EJ, Jenkins MA, Joshi AD, Joshu CE, Keku TO, Key TJ, Kim HR, Kobayashi E, Kolonel LN, Kooperberg C, Kuhn T, Kury S, Kweon SS, Larsson SC, Laurie CA, Le Marchand L, Leal SM, Lee SC, Lejbkowicz F, Lemire M, Li CI, Li L, Lieb W, Lin Y, Lindblom A, Lindor NM, Ling H, Louie TL, Mannisto S, Markowitz SD, Martin V, Masala G, McNeil CE, Melas M, Milne RL, Moreno L, Murphy N, Myte R, Naccarati A, Newcomb PA, Offit K, Ogino S, Onland-Moret NC, Pardini B, Parfrey PS, Pearlman R, Perduca V, Pharoah PDP, Pinchev M, Platz EA, Prentice RL, Pugh E, Raskin L, Rennert G, Rennert HS, Riboli E, Rodriguez-Barranco M, Romm J, Sakoda LC, Schafmayer C, Schoen RE, Seminara D, Shah M, Shelford T, Shin MH, Shulman K, Sieri S, Slattery ML, Southey MC, Stadler ZK, Stegmaier C, Su YR, Tangen CM, Thibodeau SN, Thomas DC, Thomas SS, Toland AE, Trichopoulou A, Ulrich CM, Van Den Berg DJ, van Duijnhoven FJB, Van Guelpen B, van Kranen H, Vijai J, Visvanathan K, Vodicka P, Vodickova L, Vymetalkova V, Weigl K, Weinstein SJ, White E, Win AK, Wolf CR, Wolk A, Woods MO, Wu AH, Zaidi SH, Zanke BW, Zhang Q, Zheng W, Scacheri PC, Potter JD, Bassik MC, Kundaje A, Casey G, Moreno V, Abecasis GR, Nickerson DA, Gruber SB, Hsu L, Peters U. Discovery of common and rare genetic risk variants for colorectal cancer. Nat Genet. 2019 Jan;51(1):76-87. doi: 10.1038/s41588-018-0286-6. Epub 2018 Dec 3. PMID 30510241
- [Result] Himbert C, Ose J, Nattenmuller J, Warby CA, Holowatyj AN, Bohm J, Lin T, Haffa M, Gigic B, Hardikar S, Scherer D, Zielske L, Schrotz-King P, Kolsch T, Siegel EM, Shibata D, Ulrich A, Schneider M, Hursting SD, Kauczor HU, Ulrich CM. Body Fatness, Adipose Tissue Compartments, and Biomarkers of Inflammation and Angiogenesis in Colorectal Cancer: The ColoCare Study. Cancer Epidemiol Biomarkers Prev. 2019 Jan;28(1):76-82. doi: 10.1158/1055-9965.EPI-18-0654. Epub 2018 Oct 17. PMID 30333223
- [Result] Luebeck GE, Hazelton WD, Curtius K, Maden SK, Yu M, Carter KT, Burke W, Lampe PD, Li CI, Ulrich CM, Newcomb PA, Westerhoff M, Kaz AM, Luo Y, Inadomi JM, Grady WM. Implications of Epigenetic Drift in Colorectal Neoplasia. Cancer Res. 2019 Feb 1;79(3):495-504. doi: 10.1158/0008-5472.CAN-18-1682. Epub 2018 Oct 5. PMID 30291105
- [Result] Wirbel J, Pyl PT, Kartal E, Zych K, Kashani A, Milanese A, Fleck JS, Voigt AY, Palleja A, Ponnudurai R, Sunagawa S, Coelho LP, Schrotz-King P, Vogtmann E, Habermann N, Nimeus E, Thomas AM, Manghi P, Gandini S, Serrano D, Mizutani S, Shiroma H, Shiba S, Shibata T, Yachida S, Yamada T, Waldron L, Naccarati A, Segata N, Sinha R, Ulrich CM, Brenner H, Arumugam M, Bork P, Zeller G. Meta-analysis of fecal metagenomes reveals global microbial signatures that are specific for colorectal cancer. Nat Med. 2019 Apr;25(4):679-689. doi: 10.1038/s41591-019-0406-6. Epub 2019 Apr 1. PMID 30936547
- [Result] Thomas AM, Manghi P, Asnicar F, Pasolli E, Armanini F, Zolfo M, Beghini F, Manara S, Karcher N, Pozzi C, Gandini S, Serrano D, Tarallo S, Francavilla A, Gallo G, Trompetto M, Ferrero G, Mizutani S, Shiroma H, Shiba S, Shibata T, Yachida S, Yamada T, Wirbel J, Schrotz-King P, Ulrich CM, Brenner H, Arumugam M, Bork P, Zeller G, Cordero F, Dias-Neto E, Setubal JC, Tett A, Pardini B, Rescigno M, Waldron L, Naccarati A, Segata N. Metagenomic analysis of colorectal cancer datasets identifies cross-cohort microbial diagnostic signatures and a link with choline degradation. Nat Med. 2019 Apr;25(4):667-678. doi: 10.1038/s41591-019-0405-7. Epub 2019 Apr 1. PMID 30936548
- [Result] Bien SA, Su YR, Conti DV, Harrison TA, Qu C, Guo X, Lu Y, Albanes D, Auer PL, Banbury BL, Berndt SI, Bezieau S, Brenner H, Buchanan DD, Caan BJ, Campbell PT, Carlson CS, Chan AT, Chang-Claude J, Chen S, Connolly CM, Easton DF, Feskens EJM, Gallinger S, Giles GG, Gunter MJ, Hampe J, Huyghe JR, Hoffmeister M, Hudson TJ, Jacobs EJ, Jenkins MA, Kampman E, Kang HM, Kuhn T, Kury S, Lejbkowicz F, Le Marchand L, Milne RL, Li L, Li CI, Lindblom A, Lindor NM, Martin V, McNeil CE, Melas M, Moreno V, Newcomb PA, Offit K, Pharaoh PDP, Potter JD, Qu C, Riboli E, Rennert G, Sala N, Schafmayer C, Scacheri PC, Schmit SL, Severi G, Slattery ML, Smith JD, Trichopoulou A, Tumino R, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Weinstein SJ, White E, Wolk A, Woods MO, Wu AH, Abecasis GR, Casey G, Nickerson DA, Gruber SB, Hsu L, Zheng W, Peters U. Genetic variant predictors of gene expression provide new insight into risk of colorectal cancer. Hum Genet. 2019 Apr;138(4):307-326. doi: 10.1007/s00439-019-01989-8. Epub 2019 Feb 28. PMID 30820706
- [Result] Himbert C, Ose J, Lin T, Warby CA, Gigic B, Steindorf K, Schrotz-King P, Abbenhardt-Martin C, Zielske L, Boehm J, Ulrich CM. Inflammation- and angiogenesis-related biomarkers are correlated with cancer-related fatigue in colorectal cancer patients: Results from the ColoCare Study. Eur J Cancer Care (Engl). 2019 Jul;28(4):e13055. doi: 10.1111/ecc.13055. Epub 2019 Apr 24. PMID 31016796
- [Result] Nattenmuller J, Bohm J, Bagdassarjan A, Kulu Y, Gigic B, Schneider M, Kauczor HU, Ulrich CM, Ulrich A. CT-Quantified Adipose Tissue Distribution: Risk or Protective Factor for Complications after Rectal Cancer Surgery? Obes Facts. 2019;12(3):259-271. doi: 10.1159/000499320. Epub 2019 May 3. PMID 31055588
- [Result] Haffa M, Holowatyj AN, Kratz M, Toth R, Benner A, Gigic B, Habermann N, Schrotz-King P, Bohm J, Brenner H, Schneider M, Ulrich A, Herpel E, Schirmacher P, Straub BK, Nattenmuller J, Kauczor HU, Lin T, Ball CR, Ulrich CM, Glimm H, Scherer D. Transcriptome Profiling of Adipose Tissue Reveals Depot-Specific Metabolic Alterations Among Patients with Colorectal Cancer. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5225-5237. doi: 10.1210/jc.2019-00461. PMID 31225875
- [Result] Geijsen AJMR, van Roekel EH, van Duijnhoven FJB, Achaintre D, Bachleitner-Hofmann T, Baierl A, Bergmann MM, Boehm J, Bours MJL, Brenner H, Breukink SO, Brezina S, Chang-Claude J, Herpel E, de Wilt JHW, Gicquiau A, Gigic B, Gumpenberger T, Hansson BME, Hoffmeister M, Holowatyj AN, Karner-Hanusch J, Keski-Rahkonen P, Keulen ETP, Koole JL, Leeb G, Ose J, Schirmacher P, Schneider MA, Schrotz-King P, Stift A, Ulvik A, Vogelaar FJ, Wesselink E, van Zutphen M, Gsur A, Habermann N, Kampman E, Scalbert A, Ueland PM, Ulrich AB, Ulrich CM, Weijenberg MP, Kok DE. Plasma metabolites associated with colorectal cancer stage: Findings from an international consortium. Int J Cancer. 2020 Jun 15;146(12):3256-3266. doi: 10.1002/ijc.32666. Epub 2019 Oct 10. PMID 31495913
- [Result] Ose J, Gigic B, Lin T, Liesenfeld DB, Bohm J, Nattenmuller J, Scherer D, Zielske L, Schrotz-King P, Habermann N, Ochs-Balcom HM, Peoples AR, Hardikar S, Li CI, Shibata D, Figueiredo J, Toriola AT, Siegel EM, Schmit S, Schneider M, Ulrich A, Kauczor HU, Ulrich CM. Multiplatform Urinary Metabolomics Profiling to Discriminate Cachectic from Non-Cachectic Colorectal Cancer Patients: Pilot Results from the ColoCare Study. Metabolites. 2019 Sep 6;9(9):178. doi: 10.3390/metabo9090178. PMID 31500101
- [Result] Beyerle J, Holowatyj AN, Haffa M, Frei E, Gigic B, Schrotz-King P, Boehm J, Habermann N, Stiborova M, Scherer D, Kolsch T, Skender S, Becker N, Herpel E, Schneider M, Ulrich A, Schirmacher P, Chang-Claude J, Brenner H, Hoffmeister M, Haug U, Owen RW, Ulrich CM. Expression Patterns of Xenobiotic-Metabolizing Enzymes in Tumor and Adjacent Normal Mucosa Tissues among Patients with Colorectal Cancer: The ColoCare Study. Cancer Epidemiol Biomarkers Prev. 2020 Feb;29(2):460-469. doi: 10.1158/1055-9965.EPI-19-0449. Epub 2019 Nov 18. PMID 31740522
- [Result] Holowatyj AN, Gigic B, Herpel E, Scalbert A, Schneider M, Ulrich CM; MetaboCCC Consortium; ColoCare Study. Distinct Molecular Phenotype of Sporadic Colorectal Cancers Among Young Patients Based on Multiomics Analysis. Gastroenterology. 2020 Mar;158(4):1155-1158.e2. doi: 10.1053/j.gastro.2019.11.012. Epub 2019 Nov 13. No abstract available. PMID 31730769
- [Result] Archambault AN, Su YR, Jeon J, Thomas M, Lin Y, Conti DV, Win AK, Sakoda LC, Lansdorp-Vogelaar I, Peterse EFP, Zauber AG, Duggan D, Holowatyj AN, Huyghe JR, Brenner H, Cotterchio M, Bezieau S, Schmit SL, Edlund CK, Southey MC, MacInnis RJ, Campbell PT, Chang-Claude J, Slattery ML, Chan AT, Joshi AD, Song M, Cao Y, Woods MO, White E, Weinstein SJ, Ulrich CM, Hoffmeister M, Bien SA, Harrison TA, Hampe J, Li CI, Schafmayer C, Offit K, Pharoah PD, Moreno V, Lindblom A, Wolk A, Wu AH, Li L, Gunter MJ, Gsur A, Keku TO, Pearlman R, Bishop DT, Castellvi-Bel S, Moreira L, Vodicka P, Kampman E, Giles GG, Albanes D, Baron JA, Berndt SI, Brezina S, Buch S, Buchanan DD, Trichopoulou A, Severi G, Chirlaque MD, Sanchez MJ, Palli D, Kuhn T, Murphy N, Cross AJ, Burnett-Hartman AN, Chanock SJ, de la Chapelle A, Easton DF, Elliott F, English DR, Feskens EJM, FitzGerald LM, Goodman PJ, Hopper JL, Hudson TJ, Hunter DJ, Jacobs EJ, Joshu CE, Kury S, Markowitz SD, Milne RL, Platz EA, Rennert G, Rennert HS, Schumacher FR, Sandler RS, Seminara D, Tangen CM, Thibodeau SN, Toland AE, van Duijnhoven FJB, Visvanathan K, Vodickova L, Potter JD, Mannisto S, Weigl K, Figueiredo J, Martin V, Larsson SC, Parfrey PS, Huang WY, Lenz HJ, Castelao JE, Gago-Dominguez M, Munoz-Garzon V, Mancao C, Haiman CA, Wilkens LR, Siegel E, Barry E, Younghusband B, Van Guelpen B, Harlid S, Zeleniuch-Jacquotte A, Liang PS, Du M, Casey G, Lindor NM, Le Marchand L, Gallinger SJ, Jenkins MA, Newcomb PA, Gruber SB, Schoen RE, Hampel H, Corley DA, Hsu L, Peters U, Hayes RB. Cumulative Burden of Colorectal Cancer-Associated Genetic Variants Is More Strongly Associated With Early-Onset vs Late-Onset Cancer. Gastroenterology. 2020 Apr;158(5):1274-1286.e12. doi: 10.1053/j.gastro.2019.12.012. Epub 2019 Dec 19. PMID 31866242
- [Result] Papadimitriou N, Dimou N, Tsilidis KK, Banbury B, Martin RM, Lewis SJ, Kazmi N, Robinson TM, Albanes D, Aleksandrova K, Berndt SI, Timothy Bishop D, Brenner H, Buchanan DD, Bueno-de-Mesquita B, Campbell PT, Castellvi-Bel S, Chan AT, Chang-Claude J, Ellingjord-Dale M, Figueiredo JC, Gallinger SJ, Giles GG, Giovannucci E, Gruber SB, Gsur A, Hampe J, Hampel H, Harlid S, Harrison TA, Hoffmeister M, Hopper JL, Hsu L, Maria Huerta J, Huyghe JR, Jenkins MA, Keku TO, Kuhn T, La Vecchia C, Le Marchand L, Li CI, Li L, Lindblom A, Lindor NM, Lynch B, Markowitz SD, Masala G, May AM, Milne R, Monninkhof E, Moreno L, Moreno V, Newcomb PA, Offit K, Perduca V, Pharoah PDP, Platz EA, Potter JD, Rennert G, Riboli E, Sanchez MJ, Schmit SL, Schoen RE, Severi G, Sieri S, Slattery ML, Song M, Tangen CM, Thibodeau SN, Travis RC, Trichopoulou A, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Vodicka P, White E, Wolk A, Woods MO, Wu AH, Peters U, Gunter MJ, Murphy N. Physical activity and risks of breast and colorectal cancer: a Mendelian randomisation analysis. Nat Commun. 2020 Jan 30;11(1):597. doi: 10.1038/s41467-020-14389-8. PMID 32001714
- [Result] Kiblawi R, Holowatyj AN, Gigic B, Brezina S, Geijsen AJMR, Ose J, Lin T, Hardikar S, Himbert C, Warby CA, Bohm J, Bours MJL, van Duijnhoven FJB, Gumpenberger T, Kok DE, Koole JL, van Roekel EH, Schrotz-King P, Ulvik A, Gsur A, Habermann N, Weijenberg MP, Ueland PM, Schneider M, Ulrich A, Ulrich CM, Playdon M. One-carbon metabolites, B vitamins and associations with systemic inflammation and angiogenesis biomarkers among colorectal cancer patients: results from the ColoCare Study. Br J Nutr. 2020 May 28;123(10):1187-1200. doi: 10.1017/S0007114520000422. Epub 2020 Feb 5. PMID 32019627
- [Result] Yu M, Hazelton WD, Luebeck GE, Grady WM. Epigenetic Aging: More Than Just a Clock When It Comes to Cancer. Cancer Res. 2020 Feb 1;80(3):367-374. doi: 10.1158/0008-5472.CAN-19-0924. Epub 2019 Nov 6. PMID 31694907
- [Result] Wang T, Maden SK, Luebeck GE, Li CI, Newcomb PA, Ulrich CM, Joo JE, Buchanan DD, Milne RL, Southey MC, Carter KT, Willbanks AR, Luo Y, Yu M, Grady WM. Dysfunctional epigenetic aging of the normal colon and colorectal cancer risk. Clin Epigenetics. 2020 Jan 3;12(1):5. doi: 10.1186/s13148-019-0801-3. PMID 31900199
- [Result] Han CJ, Gigic B, Schneider M, Kulu Y, Peoples AR, Ose J, Kolsch T, Jacobsen PB, Colditz GA, Figueiredo JC, Grady WM, Li CI, Shibata D, Siegel EM, Toriola AT, Ulrich AB, Syrjala KL, Ulrich CM. Risk factors for cancer-related distress in colorectal cancer survivors: one year post surgery. J Cancer Surviv. 2020 Jun;14(3):305-315. doi: 10.1007/s11764-019-00845-y. Epub 2020 Mar 12. PMID 32166576
- [Result] Gigic B, Nattenmuller J, Schneider M, Kulu Y, Syrjala KL, Bohm J, Schrotz-King P, Brenner H, Colditz GA, Figueiredo JC, Grady WM, Li CI, Shibata D, Siegel EM, Toriola AT, Kauczor HU, Ulrich A, Ulrich CM. The Role of CT-Quantified Body Composition on Longitudinal Health-Related Quality of Life in Colorectal Cancer Patients: The Colocare Study. Nutrients. 2020 Apr 28;12(5):1247. doi: 10.3390/nu12051247. PMID 32353960
- [Result] Viskochil R, Gigic B, Lin T, Skender S, Bohm J, Schrotz-King P, Steindorf K, Owen R, Figueiredo JC, Li CI, Siegel EM, Hardikar S, Shibata D, Toriola AT, Schneider M, Ulrich A, Ulrich CM, Ose J. Associations between physical activity, sedentary behavior, and urinary oxidized guanine in colorectal cancer patients: results from the ColoCare Study. Appl Physiol Nutr Metab. 2020 Nov;45(11):1306-1309. doi: 10.1139/apnm-2019-0836. Epub 2020 Jun 22. PMID 32569481
- [Result] Ose J, Holowatyj AN, Nattenmuller J, Gigic B, Lin T, Himbert C, Habermann N, Achaintre D, Scalbert A, Keski-Rahkonen P, Bohm J, Schrotz-King P, Schneider M, Ulrich A, Kampman E, Weijenberg M, Gsur A, Ueland PM, Kauczor HU, Ulrich CM. Metabolomics profiling of visceral and abdominal subcutaneous adipose tissue in colorectal cancer patients: results from the ColoCare study. Cancer Causes Control. 2020 Aug;31(8):723-735. doi: 10.1007/s10552-020-01312-1. Epub 2020 May 19. PMID 32430684
- [Result] Seyed Khoei N, Jenab M, Murphy N, Banbury BL, Carreras-Torres R, Viallon V, Kuhn T, Bueno-de-Mesquita B, Aleksandrova K, Cross AJ, Weiderpass E, Stepien M, Bulmer A, Tjonneland A, Boutron-Ruault MC, Severi G, Carbonnel F, Katzke V, Boeing H, Bergmann MM, Trichopoulou A, Karakatsani A, Martimianaki G, Palli D, Tagliabue G, Panico S, Tumino R, Sacerdote C, Skeie G, Merino S, Bonet C, Rodriguez-Barranco M, Gil L, Chirlaque MD, Ardanaz E, Myte R, Hultdin J, Perez-Cornago A, Aune D, Tsilidis KK, Albanes D, Baron JA, Berndt SI, Bezieau S, Brenner H, Campbell PT, Casey G, Chan AT, Chang-Claude J, Chanock SJ, Cotterchio M, Gallinger S, Gruber SB, Haile RW, Hampe J, Hoffmeister M, Hopper JL, Hsu L, Huyghe JR, Jenkins MA, Joshi AD, Kampman E, Larsson SC, Le Marchand L, Li CI, Li L, Lindblom A, Lindor NM, Martin V, Moreno V, Newcomb PA, Offit K, Ogino S, Parfrey PS, Pharoah PDP, Rennert G, Sakoda LC, Schafmayer C, Schmit SL, Schoen RE, Slattery ML, Thibodeau SN, Ulrich CM, van Duijnhoven FJB, Weigl K, Weinstein SJ, White E, Wolk A, Woods MO, Wu AH, Zhang X, Ferrari P, Anton G, Peters A, Peters U, Gunter MJ, Wagner KH, Freisling H. Circulating bilirubin levels and risk of colorectal cancer: serological and Mendelian randomization analyses. BMC Med. 2020 Sep 3;18(1):229. doi: 10.1186/s12916-020-01703-w. PMID 32878631
- [Result] Holowatyj AN, Haffa M, Lin T, Scherer D, Gigic B, Ose J, Warby CA, Himbert C, Abbenhardt-Martin C, Achaintre D, Boehm J, Boucher KM, Gicquiau A, Gsur A, Habermann N, Herpel E, Kauczor HU, Keski-Rahkonen P, Kloor M, von Knebel-Doeberitz M, Kok DE, Nattenmuller J, Schirmacher P, Schneider M, Schrotz-King P, Simon T, Ueland PM, Viskochil R, Weijenberg MP, Scalbert A, Ulrich A, Bowers LW, Hursting SD, Ulrich CM. Multi-omics Analysis Reveals Adipose-tumor Crosstalk in Patients with Colorectal Cancer. Cancer Prev Res (Phila). 2020 Oct;13(10):817-828. doi: 10.1158/1940-6207.CAPR-19-0538. Epub 2020 Jul 12. PMID 32655010
- [Result] Deutelmoser H, Lorenzo Bermejo J, Benner A, Weigl K, Park HA, Haffa M, Herpel E, Schneider M, Ulrich CM, Hoffmeister M, Chang-Claude J, Brenner H, Scherer D. Genotype-Based Gene Expression in Colon Tissue-Prediction Accuracy and Relationship with the Prognosis of Colorectal Cancer Patients. Int J Mol Sci. 2020 Oct 31;21(21):8150. doi: 10.3390/ijms21218150. PMID 33142733
- [Result] Wong DL, Hendrick LE, Guerrero WM, Monroe JJ, Hinkle NM, Deneve JL, Dickson PV, Glazer ES, Shibata D. Adherence to neoadjuvant therapy guidelines for locally advanced rectal cancers in a region with sociodemographic disparities. Am J Surg. 2021 Aug;222(2):395-401. doi: 10.1016/j.amjsurg.2020.11.049. Epub 2020 Nov 28. PMID 33279169
- [Result] Nounu A, Greenhough A, Heesom KJ, Richmond RC, Zheng J, Weinstein SJ, Albanes D, Baron JA, Hopper JL, Figueiredo JC, Newcomb PA, Lindor NM, Casey G, Platz EA, Le Marchand L, Ulrich CM, Li CI, van Duijnhoven FJB, Gsur A, Campbell PT, Moreno V, Vodicka P, Vodickova L, Brenner H, Chang-Claude J, Hoffmeister M, Sakoda LC, Slattery ML, Schoen RE, Gunter MJ, Castellvi-Bel S, Kim HR, Kweon SS, Chan AT, Li L, Zheng W, Bishop DT, Buchanan DD, Giles GG, Gruber SB, Rennert G, Stadler ZK, Harrison TA, Lin Y, Keku TO, Woods MO, Schafmayer C, Van Guelpen B, Gallinger S, Hampel H, Berndt SI, Pharoah PDP, Lindblom A, Wolk A, Wu AH, White E, Peters U, Drew DA, Scherer D, Bermejo JL, Williams AC, Relton CL. A Combined Proteomics and Mendelian Randomization Approach to Investigate the Effects of Aspirin-Targeted Proteins on Colorectal Cancer. Cancer Epidemiol Biomarkers Prev. 2021 Mar;30(3):564-575. doi: 10.1158/1055-9965.EPI-20-1176. Epub 2020 Dec 14. PMID 33318029
- [Result] Neumeyer S, Hua X, Seibold P, Jansen L, Benner A, Burwinkel B, Halama N, Berndt SI, Phipps AI, Sakoda LC, Schoen RE, Slattery ML, Chan AT, Gala M, Joshi AD, Ogino S, Song M, Herpel E, Blaker H, Kloor M, Scherer D, Ulrich A, Ulrich CM, Win AK, Figueiredo JC, Hopper JL, Macrae F, Milne RL, Giles GG, Buchanan DD, Peters U, Hoffmeister M, Brenner H, Newcomb PA, Chang-Claude J. Genetic Variants in the Regulatory T cell-Related Pathway and Colorectal Cancer Prognosis. Cancer Epidemiol Biomarkers Prev. 2020 Dec;29(12):2719-2728. doi: 10.1158/1055-9965.EPI-20-0714. Epub 2020 Oct 2. PMID 33008876
- [Result] Bull CJ, Bell JA, Murphy N, Sanderson E, Davey Smith G, Timpson NJ, Banbury BL, Albanes D, Berndt SI, Bezieau S, Bishop DT, Brenner H, Buchanan DD, Burnett-Hartman A, Casey G, Castellvi-Bel S, Chan AT, Chang-Claude J, Cross AJ, de la Chapelle A, Figueiredo JC, Gallinger SJ, Gapstur SM, Giles GG, Gruber SB, Gsur A, Hampe J, Hampel H, Harrison TA, Hoffmeister M, Hsu L, Huang WY, Huyghe JR, Jenkins MA, Joshu CE, Keku TO, Kuhn T, Kweon SS, Le Marchand L, Li CI, Li L, Lindblom A, Martin V, May AM, Milne RL, Moreno V, Newcomb PA, Offit K, Ogino S, Phipps AI, Platz EA, Potter JD, Qu C, Quiros JR, Rennert G, Riboli E, Sakoda LC, Schafmayer C, Schoen RE, Slattery ML, Tangen CM, Tsilidis KK, Ulrich CM, van Duijnhoven FJB, van Guelpen B, Visvanathan K, Vodicka P, Vodickova L, Wang H, White E, Wolk A, Woods MO, Wu AH, Campbell PT, Zheng W, Peters U, Vincent EE, Gunter MJ. Adiposity, metabolites, and colorectal cancer risk: Mendelian randomization study. BMC Med. 2020 Dec 17;18(1):396. doi: 10.1186/s12916-020-01855-9. PMID 33327948
- [Result] Campbell PT, Lin Y, Bien SA, Figueiredo JC, Harrison TA, Guinter MA, Berndt SI, Brenner H, Chan AT, Chang-Claude J, Gallinger SJ, Gapstur SM, Giles GG, Giovannucci E, Gruber SB, Gunter M, Hoffmeister M, Jacobs EJ, Jenkins MA, Le Marchand L, Li L, McLaughlin JR, Murphy N, Milne RL, Newcomb PA, Newton C, Ogino S, Potter JD, Rennert G, Rennert HS, Robinson J, Sakoda LC, Slattery ML, Song Y, White E, Woods MO, Casey G, Hsu L, Peters U. Association of Body Mass Index With Colorectal Cancer Risk by Genome-Wide Variants. J Natl Cancer Inst. 2021 Jan 4;113(1):38-47. doi: 10.1093/jnci/djaa058. PMID 32324875
- [Result] Brouwer JGM, Newcomb PA, Bisseling TM, Figueiredo JC, Hopper JL, Jenkins MA, Koornstra JJ, Lindor NM, Vasen HFA, Win AK, Kampman E, van Duijnhoven FJB. Associations of Height With the Risks of Colorectal and Endometrial Cancer in Persons With Lynch Syndrome. Am J Epidemiol. 2021 Feb 1;190(2):230-238. doi: 10.1093/aje/kwaa175. PMID 33524116
- [Result] Geijsen AJMR, Kok DE, van Zutphen M, Keski-Rahkonen P, Achaintre D, Gicquiau A, Gsur A, Kruyt FM, Ulrich CM, Weijenberg MP, de Wilt JHW, Wesselink E, Scalbert A, Kampman E, van Duijnhoven FJB. Diet quality indices and dietary patterns are associated with plasma metabolites in colorectal cancer patients. Eur J Nutr. 2021 Sep;60(6):3171-3184. doi: 10.1007/s00394-021-02488-1. Epub 2021 Feb 5. PMID 33544207
- [Result] Gumpenberger T, Brezina S, Keski-Rahkonen P, Baierl A, Robinot N, Leeb G, Habermann N, Kok DEG, Scalbert A, Ueland PM, Ulrich CM, Gsur A. Untargeted Metabolomics Reveals Major Differences in the Plasma Metabolome between Colorectal Cancer and Colorectal Adenomas. Metabolites. 2021 Feb 19;11(2):119. doi: 10.3390/metabo11020119. PMID 33669644
- [Result] Ose J, Gigic B, Brezina S, Lin T, Baierl A, Geijsen AJMR, van Roekel E, Robinot N, Gicquiau A, Achaintre D, Keski-Rahkonen P, Duijnhoven FJBV, Gumpenberger T, Holowatyj AN, Kok DE, Koole A, Schrotz-King P, Ulrich AB, Schneider M, Ulvik A, Ueland PM, Weijenberg MP, Habermann N, Scalbert A, Gsur A, M Ulrich C. Targeted Plasma Metabolic Profiles and Risk of Recurrence in Stage II and III Colorectal Cancer Patients: Results from an International Cohort Consortium. Metabolites. 2021 Feb 24;11(3):129. doi: 10.3390/metabo11030129. PMID 33668370
- [Result] Eisele Y, Mallea PM, Gigic B, Stephens WZ, Warby CA, Buhrke K, Lin T, Boehm J, Schrotz-King P, Hardikar S, Huang LC, Pickron TB, Scaife CL, Viskochil R, Koelsch T, Peoples AR, Pletneva MA, Bronner M, Schneider M, Ulrich AB, Swanson EA, Toriola AT, Shibata D, Li CI, Siegel EM, Figueiredo J, Janssen KP, Hauner H, Round J, Ulrich CM, Holowatyj AN, Ose J. Fusobacterium nucleatum and Clinicopathologic Features of Colorectal Cancer: Results From the ColoCare Study. Clin Colorectal Cancer. 2021 Sep;20(3):e165-e172. doi: 10.1016/j.clcc.2021.02.007. Epub 2021 Feb 27. PMID 33935016
- [Result] National Cancer Institute's PROSPR Consortium; Corley DA, Sedki M, Ritzwoller DP, Greenlee RT, Neslund-Dudas C, Rendle KA, Honda SA, Schottinger JE, Udaltsova N, Vachani A, Kobrin S, Li CI, Haas JS. Cancer Screening During the Coronavirus Disease-2019 Pandemic: A Perspective From the National Cancer Institute's PROSPR Consortium. Gastroenterology. 2021 Mar;160(4):999-1002. doi: 10.1053/j.gastro.2020.10.030. Epub 2020 Oct 21. No abstract available. PMID 33096099
- [Result] Guo X, Lin W, Wen W, Huyghe J, Bien S, Cai Q, Harrison T, Chen Z, Qu C, Bao J, Long J, Yuan Y, Wang F, Bai M, Abecasis GR, Albanes D, Berndt SI, Bezieau S, Bishop DT, Brenner H, Buch S, Burnett-Hartman A, Campbell PT, Castellvi-Bel S, Chan AT, Chang-Claude J, Chanock SJ, Cho SH, Conti DV, Chapelle A, Feskens EJM, Gallinger SJ, Giles GG, Goodman PJ, Gsur A, Guinter M, Gunter MJ, Hampe J, Hampel H, Hayes RB, Hoffmeister M, Kampman E, Kang HM, Keku TO, Kim HR, Le Marchand L, Lee SC, Li CI, Li L, Lindblom A, Lindor N, Milne RL, Moreno V, Murphy N, Newcomb PA, Nickerson DA, Offit K, Pearlman R, Pharoah PDP, Platz EA, Potter JD, Rennert G, Sakoda LC, Schafmayer C, Schmit SL, Schoen RE, Schumacher FR, Slattery ML, Su YR, Tangen CM, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Visvanathan K, Vodicka P, Vodickova L, Vymetalkova V, Wang X, White E, Wolk A, Woods MO, Casey G, Hsu L, Jenkins MA, Gruber SB, Peters U, Zheng W. Identifying Novel Susceptibility Genes for Colorectal Cancer Risk From a Transcriptome-Wide Association Study of 125,478 Subjects. Gastroenterology. 2021 Mar;160(4):1164-1178.e6. doi: 10.1053/j.gastro.2020.08.062. Epub 2020 Oct 12. PMID 33058866
- [Result] Schmitt FCF, Schneider M, Mathejczyk W, Weigand MA, Figueiredo JC, Li CI, Shibata D, Siegel EM, Toriola AT, Ulrich CM, Ulrich AB, Boutin S, Gigic B. Postoperative Complications Are Associated with Long-Term Changes in the Gut Microbiota Following Colorectal Cancer Surgery. Life (Basel). 2021 Mar 16;11(3):246. doi: 10.3390/life11030246. PMID 33809741
- [Result] Matejcic M, Shaban HA, Quintana MW, Schumacher FR, Edlund CK, Naghi L, Pai RK, Haile RW, Levine AJ, Buchanan DD, Jenkins MA, Figueiredo JC, Rennert G, Gruber SB, Li L, Casey G, Conti DV, Schmit SL. Rare Variants in the DNA Repair Pathway and the Risk of Colorectal Cancer. Cancer Epidemiol Biomarkers Prev. 2021 May;30(5):895-903. doi: 10.1158/1055-9965.EPI-20-1457. Epub 2021 Feb 24. PMID 33627384
- [Result] Jenkins MA, Buchanan DD, Lai J, Makalic E, Dite GS, Win AK, Clendenning M, Winship IM, Hayes RB, Huyghe JR, Peters U, Gallinger S, Marchand LL, Figueiredo JC, Pai RK, Newcomb PA, Church JM, Casey G, Hopper JL. Assessment of a Polygenic Risk Score for Colorectal Cancer to Predict Risk of Lynch Syndrome Colorectal Cancer. JNCI Cancer Spectr. 2021 Mar 8;5(2):pkab022. doi: 10.1093/jncics/pkab022. eCollection 2021 Apr. PMID 33928216
- [Result] Benson AB, Venook AP, Al-Hawary MM, Arain MA, Chen YJ, Ciombor KK, Cohen S, Cooper HS, Deming D, Farkas L, Garrido-Laguna I, Grem JL, Gunn A, Hecht JR, Hoffe S, Hubbard J, Hunt S, Johung KL, Kirilcuk N, Krishnamurthi S, Messersmith WA, Meyerhardt J, Miller ED, Mulcahy MF, Nurkin S, Overman MJ, Parikh A, Patel H, Pedersen K, Saltz L, Schneider C, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Gregory KM, Gurski LA. Colon Cancer, Version 2.2021, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2021 Mar 2;19(3):329-359. doi: 10.6004/jnccn.2021.0012. PMID 33724754
- [Result] Biltaji E, Walker B, Au TH, Rivers Z, Ose J, Li CI, Brixner DI, Stenehjem DD, Ulrich CM. Can Cost-effectiveness Analysis Inform Genotype-Guided Aspirin Use for Primary Colorectal Cancer Prevention? Cancer Epidemiol Biomarkers Prev. 2021 Jun;30(6):1106-1113. doi: 10.1158/1055-9965.EPI-19-1580. Epub 2021 Apr 13. PMID 33849967
- [Result] Archambault AN, Lin Y, Jeon J, Harrison TA, Bishop DT, Brenner H, Casey G, Chan AT, Chang-Claude J, Figueiredo JC, Gallinger S, Gruber SB, Gunter MJ, Hoffmeister M, Jenkins MA, Keku TO, Marchand LL, Li L, Moreno V, Newcomb PA, Pai R, Parfrey PS, Rennert G, Sakoda LC, Sandler RS, Slattery ML, Song M, Win AK, Woods MO, Murphy N, Campbell PT, Su YR, Zeleniuch-Jacquotte A, Liang PS, Du M, Hsu L, Peters U, Hayes RB. Nongenetic Determinants of Risk for Early-Onset Colorectal Cancer. JNCI Cancer Spectr. 2021 May 20;5(3):pkab029. doi: 10.1093/jncics/pkab029. eCollection 2021 Jun. PMID 34041438
- [Result] Kamal Y, Dwan D, Hoehn HJ, Sanz-Pamplona R, Alonso MH, Moreno V, Cheng C, Schell MJ, Kim Y, Felder SI, Rennert HS, Melas M, Lazaris C, Bonner JD, Siegel EM, Shibata D, Rennert G, Gruber SB, Frost HR, Amos CI, Schmit SL. Tumor immune infiltration estimated from gene expression profiles predicts colorectal cancer relapse. Oncoimmunology. 2021 Mar 9;10(1):1862529. doi: 10.1080/2162402X.2020.1862529. PMID 33763292
- [Result] Pan XF, Yang JJ, Shu XO, Moore SC, Palmer ND, Guasch-Ferre M, Herrington DM, Harada S, Eliassen H, Wang TJ, Gerszten RE, Albanes D, Tzoulaki I, Karaman I, Elliott P, Zhu H, Wagenknecht LE, Zheng W, Cai H, Cai Q, Matthews CE, Menni C, Meyer KA, Lipworth LP, Ose J, Fornage M, Ulrich CM, Yu D. Associations of circulating choline and its related metabolites with cardiometabolic biomarkers: an international pooled analysis. Am J Clin Nutr. 2021 Sep 1;114(3):893-906. doi: 10.1093/ajcn/nqab152. PMID 34020444
- [Result] Koole JL, Bours MJL, Geijsen AJMR, Gigic B, Ulvik A, Kok DE, Brezina S, Ose J, Baierl A, Bohm J, Brenner H, Breukink SO, Chang-Claude J, van Duijnhoven FJB, van Duijvendijk P, Gumpenberger T, Habermann N, van Halteren HK, Hoffmeister M, Holowatyj AN, Janssen-Heijnen MLG, Keulen ETP, Kiblawi R, Kruyt FM, Li CI, Lin T, Midttun O, Peoples AR, van Roekel EH, Schneider MA, Schrotz-King P, Ulrich AB, Vickers K, Wesselink E, de Wilt JHW, Gsur A, Ueland PM, Ulrich CM, Kampman E, Weijenberg MP. Circulating B-vitamin biomarkers and B-vitamin supplement use in relation to quality of life in patients with colorectal cancer: results from the FOCUS consortium. Am J Clin Nutr. 2021 Jun 1;113(6):1468-1481. doi: 10.1093/ajcn/nqaa422. PMID 33668069
- [Result] Tsilidis KK, Papadimitriou N, Dimou N, Gill D, Lewis SJ, Martin RM, Murphy N, Markozannes G, Zuber V, Cross AJ, Burrows K, Lopez DS, Key TJ, Travis RC, Perez-Cornago A, Hunter DJ, van Duijnhoven FJB, Albanes D, Arndt V, Berndt SI, Bezieau S, Bishop DT, Boehm J, Brenner H, Burnett-Hartman A, Campbell PT, Casey G, Castellvi-Bel S, Chan AT, Chang-Claude J, de la Chapelle A, Figueiredo JC, Gallinger SJ, Giles GG, Goodman PJ, Gsur A, Hampe J, Hampel H, Hoffmeister M, Jenkins MA, Keku TO, Kweon SS, Larsson SC, Le Marchand L, Li CI, Li L, Lindblom A, Martin V, Milne RL, Moreno V, Nan H, Nassir R, Newcomb PA, Offit K, Pharoah PDP, Platz EA, Potter JD, Qi L, Rennert G, Sakoda LC, Schafmayer C, Slattery ML, Snetselaar L, Schenk J, Thibodeau SN, Ulrich CM, Van Guelpen B, Harlid S, Visvanathan K, Vodickova L, Wang H, White E, Wolk A, Woods MO, Wu AH, Zheng W, Bueno-de-Mesquita B, Boutron-Ruault MC, Hughes DJ, Jakszyn P, Kuhn T, Palli D, Riboli E, Giovannucci EL, Banbury BL, Gruber SB, Peters U, Gunter MJ. Genetically predicted circulating concentrations of micronutrients and risk of colorectal cancer among individuals of European descent: a Mendelian randomization study. Am J Clin Nutr. 2021 Jun 1;113(6):1490-1502. doi: 10.1093/ajcn/nqab003. PMID 33740060
- [Result] Hathaway CA, Chavez MN, Kadono M, Ketcher D, Rollison DE, Siegel EM, Peoples AR, Ulrich CM, Penedo FJ, Tworoger SS, Gonzalez BD. Improving Electronic Survey Response Rates Among Cancer Center Patients During the COVID-19 Pandemic: Mixed Methods Pilot Study. JMIR Cancer. 2021 Aug 6;7(3):e30265. doi: 10.2196/30265. PMID 34156965
- [Result] Papadimitriou N, Gunter MJ, Murphy N, Gicquiau A, Achaintre D, Brezina S, Gumpenberger T, Baierl A, Ose J, Geijsen AJMR, van Roekel EH, Gsur A, Gigic B, Habermann N, Ulrich CM, Kampman E, Weijenberg MP, Ueland PM, Kaaks R, Katzke V, Krogh V, Bueno-de-Mesquita B, Ardanaz E, Travis RC, Schulze MB, Sanchez MJ, Colorado-Yohar SM, Weiderpass E, Scalbert A, Keski-Rahkonen P. Circulating tryptophan metabolites and risk of colon cancer: Results from case-control and prospective cohort studies. Int J Cancer. 2021 Nov 1;149(9):1659-1669. doi: 10.1002/ijc.33725. Epub 2021 Jul 12. PMID 34196970
- [Result] Figueiredo JC, Jacobs EJ, Newton CC, Guinter MA, Cance WG, Campbell PT. Associations of Aspirin and Non-Aspirin Non-Steroidal Anti-Inflammatory Drugs With Colorectal Cancer Mortality After Diagnosis. J Natl Cancer Inst. 2021 Jul 1;113(7):833-840. doi: 10.1093/jnci/djab008. PMID 33528005
- [Result] Deschner BW, VanderWalde NA, Grothey A, Shibata D. Evolution and Current Status of the Multidisciplinary Management of Locally Advanced Rectal Cancer. JCO Oncol Pract. 2021 Jul;17(7):383-402. doi: 10.1200/OP.20.00885. Epub 2021 Apr 21. PMID 33881906
- [Result] Huyghe JR, Harrison TA, Bien SA, Hampel H, Figueiredo JC, Schmit SL, Conti DV, Chen S, Qu C, Lin Y, Barfield R, Baron JA, Cross AJ, Diergaarde B, Duggan D, Harlid S, Imaz L, Kang HM, Levine DM, Perduca V, Perez-Cornago A, Sakoda LC, Schumacher FR, Slattery ML, Toland AE, van Duijnhoven FJB, Van Guelpen B, Agudo A, Albanes D, Alonso MH, Anderson K, Arnau-Collell C, Arndt V, Banbury BL, Bassik MC, Berndt SI, Bezieau S, Bishop DT, Boehm J, Boeing H, Boutron-Ruault MC, Brenner H, Brezina S, Buch S, Buchanan DD, Burnett-Hartman A, Caan BJ, Campbell PT, Carr PR, Castells A, Castellvi-Bel S, Chan AT, Chang-Claude J, Chanock SJ, Curtis KR, de la Chapelle A, Easton DF, English DR, Feskens EJM, Gala M, Gallinger SJ, Gauderman WJ, Giles GG, Goodman PJ, Grady WM, Grove JS, Gsur A, Gunter MJ, Haile RW, Hampe J, Hoffmeister M, Hopper JL, Hsu WL, Huang WY, Hudson TJ, Jenab M, Jenkins MA, Joshi AD, Keku TO, Kooperberg C, Kuhn T, Kury S, Le Marchand L, Lejbkowicz F, Li CI, Li L, Lieb W, Lindblom A, Lindor NM, Mannisto S, Markowitz SD, Milne RL, Moreno L, Murphy N, Nassir R, Offit K, Ogino S, Panico S, Parfrey PS, Pearlman R, Pharoah PDP, Phipps AI, Platz EA, Potter JD, Prentice RL, Qi L, Raskin L, Rennert G, Rennert HS, Riboli E, Schafmayer C, Schoen RE, Seminara D, Song M, Su YR, Tangen CM, Thibodeau SN, Thomas DC, Trichopoulou A, Ulrich CM, Visvanathan K, Vodicka P, Vodickova L, Vymetalkova V, Weigl K, Weinstein SJ, White E, Wolk A, Woods MO, Wu AH, Abecasis GR, Nickerson DA, Scacheri PC, Kundaje A, Casey G, Gruber SB, Hsu L, Moreno V, Hayes RB, Newcomb PA, Peters U. Genetic architectures of proximal and distal colorectal cancer are partly distinct. Gut. 2021 Jul;70(7):1325-1334. doi: 10.1136/gutjnl-2020-321534. Epub 2021 Feb 25. PMID 33632709
- [Result] Himbert C, Hathaway CA, Daniels B, Salas K, Ashworth A, Gigic B, Lin T, Viskochil R, Kirchhoff AC, Grossman D, Ose J, Tward J, Scaife C, Figueiredo JC, Toriola AT, Beck A, Shibata D, Gonzalez BD, Matsen C, Christenson C, Ma DS, Colman H, Hunt JP, Jones KB, Lee CJ, Larson M, Onega T, Akerley WL, Li CI, Schneider M, Penedo FJ, Siegel EM, Tworoger SS, Ulrich CM, Peoples AR. Impact of the COVID-19 pandemic on exercise habits among cancer patients. Res Sq [Preprint]. 2021 Sep 21:rs.3.rs-704646. doi: 10.21203/rs.3.rs-704646/v1. PMID 34580667
- [Result] Lindley CL, Gigic B, Peoples AR, Han CJ, Lin T, Himbert C, Warby CA, Boehm J, Hardikar S, Ashworth A, Schneider M, Ulrich A, Schrotz-King P, Figueiredo JC, Li CI, Shibata D, Siegel EM, Toriola AT, Ulrich CM, Syrjala KL, Ose J. Pre-Surgery Inflammatory and Angiogenesis Biomarkers as Predictors of 12-Month Cancer-Related Distress: Results from the ColoCare Study. Cancer Epidemiol Biomarkers Prev. 2023 Mar 6;32(3):363-370. doi: 10.1158/1055-9965.EPI-22-0882. PMID 36595657
- [Result] Carreras-Torres R, Kim AE, Lin Y, Diez-Obrero V, Bien SA, Qu C, Wang J, Dimou N, Aglago EK, Albanes D, Arndt V, Baurley JW, Berndt SI, Bezieau S, Bishop DT, Bouras E, Brenner H, Budiarto A, Campbell PT, Casey G, Chan AT, Chang-Claude J, Chen X, Conti DV, Dampier CH, Devall MAM, Drew DA, Figueiredo JC, Gallinger S, Giles GG, Gruber SB, Gsur A, Gunter MJ, Harrison TA, Hidaka A, Hoffmeister M, Huyghe JR, Jenkins MA, Jordahl KM, Kawaguchi E, Keku TO, Kundaje A, Le Marchand L, Lewinger JP, Li L, Mahesworo B, Morrison JL, Murphy N, Nan H, Nassir R, Newcomb PA, Obon-Santacana M, Ogino S, Ose J, Pai RK, Palmer JR, Papadimitriou N, Pardamean B, Peoples AR, Pharoah PDP, Platz EA, Rennert G, Ruiz-Narvaez E, Sakoda LC, Scacheri PC, Schmit SL, Schoen RE, Shcherbina A, Slattery ML, Stern MC, Su YR, Tangen CM, Thomas DC, Tian Y, Tsilidis KK, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Visvanathan K, Vodicka P, Cenggoro TW, Weinstein SJ, White E, Wolk A, Woods MO, Hsu L, Peters U, Moreno V, Gauderman WJ. Genome-wide Interaction Study with Smoking for Colorectal Cancer Risk Identifies Novel Genetic Loci Related to Tumor Suppression, Inflammation, and Immune Response. Cancer Epidemiol Biomarkers Prev. 2023 Mar 6;32(3):315-328. doi: 10.1158/1055-9965.EPI-22-0763. PMID 36576985
- [Result] Papadimitriou N, Bull CJ, Jenab M, Hughes DJ, Bell JA, Sanderson E, Timpson NJ, Smith GD, Albanes D, Campbell PT, Kury S, Le Marchand L, Ulrich CM, Visvanathan K, Figueiredo JC, Newcomb PA, Pai RK, Peters U, Tsilidis KK, Boer JMA, Vincent EE, Mariosa D, Gunter MJ, Richardson TG, Murphy N. Separating the effects of early and later life adiposity on colorectal cancer risk: a Mendelian randomization study. BMC Med. 2023 Jan 4;21(1):5. doi: 10.1186/s12916-022-02702-9. PMID 36600297
- [Result] Thomas M, Su YR, Rosenthal EA, Sakoda LC, Schmit SL, Timofeeva MN, Chen Z, Fernandez-Rozadilla C, Law PJ, Murphy N, Carreras-Torres R, Diez-Obrero V, van Duijnhoven FJ, Jiang S, Shin A, Wolk A, Phipps AI, Burnett-Hartman A, Gsur A, Chan AT, Zauber AG, Wu AH, Lindblom A, Um CY, Tangen CM, Gignoux C, Newton C, Haiman CA, Qu C, Bishop DT, Buchanan DD, Crosslin DR, Conti DV, Kim DH, Hauser E, White E, Siegel E, Schumacher FR, Rennert G, Giles GG, Hampel H, Brenner H, Oze I, Oh JH, Lee JK, Schneider JL, Chang-Claude J, Kim J, Huyghe JR, Zheng J, Hampe J, Greenson J, Hopper JL, Palmer JR, Visvanathan K, Matsuo K, Matsuda K, Jung KJ, Li L, Marchand LL, Vodickova L, Bujanda L, Gunter MJ, Matejcic M, Jenkins MA, Slattery ML, D'Amato M, Wang M, Hoffmeister M, Woods MO, Kim M, Song M, Iwasaki M, Du M, Udaltsova N, Sawada N, Vodicka P, Campbell PT, Newcomb PA, Cai Q, Pearlman R, Pai RK, Schoen RE, Steinfelder RS, Haile RW, Vandenputtelaar R, Prentice RL, Kury S, Castellvi-Bel S, Tsugane S, Berndt SI, Lee SC, Brezina S, Weinstein SJ, Chanock SJ, Jee SH, Kweon SS, Vadaparampil S, Harrison TA, Yamaji T, Keku TO, Vymetalkova V, Arndt V, Jia WH, Shu XO, Lin Y, Ahn YO, Stadler ZK, Van Guelpen B, Ulrich CM, Platz EA, Potter JD, Li CI, Meester R, Moreno V, Figueiredo JC, Casey G, Vogelaar IL, Dunlop MG, Gruber SB, Hayes RB, Pharoah PDP, Houlston RS, Jarvik GP, Tomlinson IP, Zheng W, Corley DA, Peters U, Hsu L. Combining Asian-European Genome-Wide Association Studies of Colorectal Cancer Improves Risk Prediction Across Race and Ethnicity. medRxiv [Preprint]. 2023 Jan 19:2023.01.19.23284737. doi: 10.1101/2023.01.19.23284737. PMID 36789420
- [Result] Berghuijs KMVT, Kaddas HK, Trujillo G, Rouhani G, Chevrier A, Ose J, Shibata D, Toriola AT, Figueiredo JC, Peoples AR, Li CI, Hardikar S, Siegel EM, Gigic B, Schneider M, Ulrich CM, Kirchhoff AC. Age-related differences in employment, insurance, and financial hardship among colorectal cancer patients: a report from the ColoCare Study. J Cancer Surviv. 2024 Jun;18(3):1075-1084. doi: 10.1007/s11764-023-01362-9. Epub 2023 Mar 23. PMID 36949233
- [Result] Cheng TD, Ilozumba MN, Balavarca Y, Neuhouser ML, Miller JW, Beresford SAA, Zheng Y, Song X, Duggan DJ, Toriola AT, Bailey LB, Green R, Caudill MA, Ulrich CM. Associations between Genetic Variants and Blood Biomarkers of One-Carbon Metabolism in Postmenopausal Women from the Women's Health Initiative Observational Study. J Nutr. 2022 Apr 1;152(4):1099-1106. doi: 10.1093/jn/nxab444. PMID 34967850
- [Result] Himbert C, Ose J, Gigic B, Viskochil R, Santuci K, Lin T, Ashworth A, Cohan JN, Scaife CL, Jedrzkiewicz J, Damerell V, Atkins KM, Gong J, Mutch MG, Bernadt C, Felder S, Sanchez J, Cohen SA, Krane MK, Hinkle N, Wood E, Peoples AR, Figueiredo JC, Toriola AT, Siegel EM, Li CI, Shibata D, Boucher K, Round JL, Ulrich AB, Schneider M, Huang LC, Hardikar S, Ulrich CM. Associations of combined physical activity and body mass index groups with colorectal cancer survival outcomes. BMC Cancer. 2023 Apr 3;23(1):300. doi: 10.1186/s12885-023-10695-8. PMID 37013476
- [Result] Aglago EK, Kim A, Lin Y, Qu C, Evangelou M, Ren Y, Morrison J, Albanes D, Arndt V, Barry EL, Baurley JW, Berndt SI, Bien SA, Bishop DT, Bouras E, Brenner H, Buchanan DD, Budiarto A, Carreras-Torres R, Casey G, Cenggoro TW, Chan AT, Chang-Claude J, Chen X, Conti DV, Devall M, Diez-Obrero V, Dimou N, Drew D, Figueiredo JC, Gallinger S, Giles GG, Gruber SB, Gsur A, Gunter MJ, Hampel H, Harlid S, Hidaka A, Harrison TA, Hoffmeister M, Huyghe JR, Jenkins MA, Jordahl K, Joshi AD, Kawaguchi ES, Keku TO, Kundaje A, Larsson SC, Marchand LL, Lewinger JP, Li L, Lynch BM, Mahesworo B, Mandic M, Obon-Santacana M, Moreno V, Murphy N, Nan H, Nassir R, Newcomb PA, Ogino S, Ose J, Pai RK, Palmer JR, Papadimitriou N, Pardamean B, Peoples AR, Platz EA, Potter JD, Prentice RL, Rennert G, Ruiz-Narvaez E, Sakoda LC, Scacheri PC, Schmit SL, Schoen RE, Shcherbina A, Slattery ML, Stern MC, Su YR, Tangen CM, Thibodeau SN, Thomas DC, Tian Y, Ulrich CM, van Duijnhoven FJ, Van Guelpen B, Visvanathan K, Vodicka P, Wang J, White E, Wolk A, Woods MO, Wu AH, Zemlianskaia N, Hsu L, Gauderman WJ, Peters U, Tsilidis KK, Campbell PT. A Genetic Locus within the FMN1/GREM1 Gene Region Interacts with Body Mass Index in Colorectal Cancer Risk. Cancer Res. 2023 Aug 1;83(15):2572-2583. doi: 10.1158/0008-5472.CAN-22-3713. PMID 37249599
- [Result] Wheeler CE, Coleman SS 4th, Hoyd R, Denko L, Chan CHF, Churchman ML, Denko N, Dodd RD, Eljilany I, Hardikar S, Husain M, Ikeguchi AP, Jin N, Ma Q, McCarter MD, Osman AEG, Robinson LA, Singer EA, Tinoco G, Ulrich CM, Zakharia Y, Spakowicz D, Tarhini AA, Tan AC. The tumor microbiome as a predictor of outcomes in patients with metastatic melanoma treated with immune checkpoint inhibitors. bioRxiv [Preprint]. 2023 May 25:2023.05.24.542123. doi: 10.1101/2023.05.24.542123. PMID 37292921
- [Result] Wang C, Ma A, McNutt ME, Hoyd R, Wheeler CE, Robinson LA, Chan CHF, Zakharia Y, Dodd RD, Ulrich CM, Hardikar S, Churchman ML, Tarhini AA, Singer EA, Ikeguchi AP, McCarter MD, Denko N, Tinoco G, Husain M, Jin N, Osman AEG, Eljilany I, Tan AC, Coleman SS 4th, Denko L, Riedlinger G, Schneider BP, Spakowicz D, Ma Q. A bioinformatics tool for identifying intratumoral microbes from the ORIEN dataset. bioRxiv [Preprint]. 2023 May 24:2023.05.24.541982. doi: 10.1101/2023.05.24.541982. PMID 37292990
- [Result] Yu M, Carter KT, Baker KK, Redman MW, Wang T, Vickers K, Li CI, Cohen SA, Krane M, Ose J, Gigic B, Figueiredo JC, Toriola AT, Siegel EM, Shibata D, Schneider M, Ulrich CM, Dzubinski LA, Schoen RE, Grady WM. Elevated EVL Methylation Level in the Normal Colon Mucosa Is a Potential Risk Biomarker for Developing Recurrent Adenomas. Cancer Epidemiol Biomarkers Prev. 2023 Sep 1;32(9):1146-1152. doi: 10.1158/1055-9965.EPI-22-1020. PMID 37294695
- [Result] Thomas M, Su YR, Rosenthal EA, Sakoda LC, Schmit SL, Timofeeva MN, Chen Z, Fernandez-Rozadilla C, Law PJ, Murphy N, Carreras-Torres R, Diez-Obrero V, van Duijnhoven FJB, Jiang S, Shin A, Wolk A, Phipps AI, Burnett-Hartman A, Gsur A, Chan AT, Zauber AG, Wu AH, Lindblom A, Um CY, Tangen CM, Gignoux C, Newton C, Haiman CA, Qu C, Bishop DT, Buchanan DD, Crosslin DR, Conti DV, Kim DH, Hauser E, White E, Siegel E, Schumacher FR, Rennert G, Giles GG, Hampel H, Brenner H, Oze I, Oh JH, Lee JK, Schneider JL, Chang-Claude J, Kim J, Huyghe JR, Zheng J, Hampe J, Greenson J, Hopper JL, Palmer JR, Visvanathan K, Matsuo K, Matsuda K, Jung KJ, Li L, Le Marchand L, Vodickova L, Bujanda L, Gunter MJ, Matejcic M, Jenkins MA, Slattery ML, D'Amato M, Wang M, Hoffmeister M, Woods MO, Kim M, Song M, Iwasaki M, Du M, Udaltsova N, Sawada N, Vodicka P, Campbell PT, Newcomb PA, Cai Q, Pearlman R, Pai RK, Schoen RE, Steinfelder RS, Haile RW, Vandenputtelaar R, Prentice RL, Kury S, Castellvi-Bel S, Tsugane S, Berndt SI, Lee SC, Brezina S, Weinstein SJ, Chanock SJ, Jee SH, Kweon SS, Vadaparampil S, Harrison TA, Yamaji T, Keku TO, Vymetalkova V, Arndt V, Jia WH, Shu XO, Lin Y, Ahn YO, Stadler ZK, Van Guelpen B, Ulrich CM, Platz EA, Potter JD, Li CI, Meester R, Moreno V, Figueiredo JC, Casey G, Lansdorp Vogelaar I, Dunlop MG, Gruber SB, Hayes RB, Pharoah PDP, Houlston RS, Jarvik GP, Tomlinson IP, Zheng W, Corley DA, Peters U, Hsu L. Combining Asian and European genome-wide association studies of colorectal cancer improves risk prediction across racial and ethnic populations. Nat Commun. 2023 Oct 2;14(1):6147. doi: 10.1038/s41467-023-41819-0. PMID 37783704
- [Result] Crowder SL, Li X, Himbert C, Viskochil R, Hoogland AI, Gudenkauf LM, Oswald LB, Gonzalez BD, Small BJ, Ulrich CM, Ose J, Peoples AR, Li CI, Shibata D, Toriola AT, Gigic B, Playdon MC, Hardikar S, Bower J, Siegel EM, Figueiredo JC, Jim HSL. Relationships Among Physical Activity, Sleep, and Cancer-related Fatigue: Results From the International ColoCare Study. Ann Behav Med. 2024 Feb 10;58(3):156-166. doi: 10.1093/abm/kaad068. PMID 38141201
- [Result] Etemad M, Christodoulou F, Uhlig S, Hassel JC, Schrotz-King P, Brenner H, Ulrich CM, Bieback K, Kluter H, Bugert P. C-Type Lectin-like Receptor 2 Expression Is Decreased upon Platelet Activation and Is Lower in Most Tumor Entities Compared to Healthy Controls. Cancers (Basel). 2023 Nov 22;15(23):5514. doi: 10.3390/cancers15235514. PMID 38067218
- [Result] Stern MC, Sanchez Mendez J, Kim AE, Obon-Santacana M, Moratalla-Navarro F, Martin V, Moreno V, Lin Y, Bien SA, Qu C, Su YR, White E, Harrison TA, Huyghe JR, Tangen CM, Newcomb PA, Phipps AI, Thomas CE, Kawaguchi ES, Lewinger JP, Morrison JL, Conti DV, Wang J, Thomas DC, Platz EA, Visvanathan K, Keku TO, Newton CC, Um CY, Kundaje A, Shcherbina A, Murphy N, Gunter MJ, Dimou N, Papadimitriou N, Bezieau S, van Duijnhoven FJB, Mannisto S, Rennert G, Wolk A, Hoffmeister M, Brenner H, Chang-Claude J, Tian Y, Le Marchand L, Cotterchio M, Tsilidis KK, Bishop DT, Melaku YA, Lynch BM, Buchanan DD, Ulrich CM, Ose J, Peoples AR, Pellatt AJ, Li L, Devall MAM, Campbell PT, Albanes D, Weinstein SJ, Berndt SI, Gruber SB, Ruiz-Narvaez E, Song M, Joshi AD, Drew DA, Petrick JL, Chan AT, Giannakis M, Peters U, Hsu L, Gauderman WJ. Genome-Wide Gene-Environment Interaction Analyses to Understand the Relationship between Red Meat and Processed Meat Intake and Colorectal Cancer Risk. Cancer Epidemiol Biomarkers Prev. 2024 Mar 1;33(3):400-410. doi: 10.1158/1055-9965.EPI-23-0717. PMID 38112776
- [Result] Kok DE, van Duijnhoven FJ, Lubberman FJ, McKay JA, Lanen AV, Winkels RM, Wesselink E, van Halteren HK, de Wilt JH, Ulrich CM, Ulvik A, Ueland PM, Kampman E. Intake and biomarkers of folate and folic acid as determinants of chemotherapy-induced toxicities in patients with colorectal cancer: a cohort study. Am J Clin Nutr. 2024 Feb;119(2):294-301. doi: 10.1016/j.ajcnut.2023.11.023. Epub 2023 Dec 7. PMID 38070682
- [Result] Li X, Hoogland AI, Small BJ, Crowder SL, Gonzalez BD, Oswald LB, Sleight AG, Nguyen N, Lorona NC, Damerell V, Komrokji KR, Mooney K, Playdon MC, Ulrich CM, Li CI, Shibata D, Toriola AT, Ose J, Peoples AR, Siegel EM, Bower JE, Schneider M, Gigic B, Figueiredo JC, Jim HSL. Trajectories and risk factors of fatigue following colorectal cancer diagnosis. Colorectal Dis. 2023 Oct;25(10):2054-2063. doi: 10.1111/codi.16746. Epub 2023 Sep 12. PMID 37700526
- [Result] Bouras E, Kim AE, Lin Y, Morrison J, Du M, Albanes D, Barry EL, Baurley JW, Berndt SI, Bien SA, Bishop TD, Brenner H, Budiarto A, Burnett-Hartman A, Campbell PT, Carreras-Torres R, Casey G, Cenggoro TW, Chan AT, Chang-Claude J, Conti DV, Cotterchio M, Devall M, Diez-Obrero V, Dimou N, Drew DA, Figueiredo JC, Giles GG, Gruber SB, Gunter MJ, Harrison TA, Hidaka A, Hoffmeister M, Huyghe JR, Joshi AD, Kawaguchi ES, Keku TO, Kundaje A, Le Marchand L, Lewinger JP, Li L, Lynch BM, Mahesworo B, Mannisto S, Moreno V, Murphy N, Newcomb PA, Obon-Santacana M, Ose J, Palmer JR, Papadimitriou N, Pardamean B, Pellatt AJ, Peoples AR, Platz EA, Potter JD, Qi L, Qu C, Rennert G, Ruiz-Narvaez E, Sakoda LC, Schmit SL, Shcherbina A, Stern MC, Su YR, Tangen CM, Thomas DC, Tian Y, Um CY, van Duijnhoven FJ, Van Guelpen B, Visvanathan K, Wang J, White E, Wolk A, Woods MO, Ulrich CM, Hsu L, Gauderman WJ, Peters U, Tsilidis KK. Genome-wide interaction analysis of folate for colorectal cancer risk. Am J Clin Nutr. 2023 Nov;118(5):881-891. doi: 10.1016/j.ajcnut.2023.08.010. Epub 2023 Aug 26. PMID 37640106
- [Result] Dimou N, Kim AE, Flanagan O, Murphy N, Diez-Obrero V, Shcherbina A, Aglago EK, Bouras E, Campbell PT, Casey G, Gallinger S, Gruber SB, Jenkins MA, Lin Y, Moreno V, Ruiz-Narvaez E, Stern MC, Tian Y, Tsilidis KK, Arndt V, Barry EL, Baurley JW, Berndt SI, Bezieau S, Bien SA, Bishop DT, Brenner H, Budiarto A, Carreras-Torres R, Cenggoro TW, Chan AT, Chang-Claude J, Chanock SJ, Chen X, Conti DV, Dampier CH, Devall M, Drew DA, Figueiredo JC, Giles GG, Gsur A, Harrison TA, Hidaka A, Hoffmeister M, Huyghe JR, Jordahl K, Kawaguchi E, Keku TO, Larsson SC, Le Marchand L, Lewinger JP, Li L, Mahesworo B, Morrison J, Newcomb PA, Newton CC, Obon-Santacana M, Ose J, Pai RK, Palmer JR, Papadimitriou N, Pardamean B, Peoples AR, Pharoah PDP, Platz EA, Potter JD, Rennert G, Scacheri PC, Schoen RE, Su YR, Tangen CM, Thibodeau SN, Thomas DC, Ulrich CM, Um CY, van Duijnhoven FJB, Visvanathan K, Vodicka P, Vodickova L, White E, Wolk A, Woods MO, Qu C, Kundaje A, Hsu L, Gauderman WJ, Gunter MJ, Peters U. Probing the diabetes and colorectal cancer relationship using gene - environment interaction analyses. Br J Cancer. 2023 Aug;129(3):511-520. doi: 10.1038/s41416-023-02312-z. Epub 2023 Jun 26. PMID 37365285
- [Result] Ose J, Gigic B, Brezina S, Lin T, Peoples AR, Schobert PP, Baierl A, van Roekel E, Robinot N, Gicquiau A, Achaintre D, Scalbert A, van Duijnhoven FJB, Holowatyj AN, Gumpenberger T, Schrotz-King P, Ulrich AB, Ulvik A, Ueland PM, Weijenberg MP, Habermann N, Keski-Rahkonen P, Gsur A, Kok DE, Ulrich CM. Higher Plasma Creatinine Is Associated with an Increased Risk of Death in Patients with Non-Metastatic Rectal but Not Colon Cancer: Results from an International Cohort Consortium. Cancers (Basel). 2023 Jun 28;15(13):3391. doi: 10.3390/cancers15133391. PMID 37444500
- [Result] Mahmood K, Thomas M, Qu C; Gecco-Ccfr Consortium; Hsu L, Buchanan DD, Peters U. Elucidating the Risk of Colorectal Cancer for Variants in Hereditary Colorectal Cancer Genes. Gastroenterology. 2023 Oct;165(4):1070-1076.e3. doi: 10.1053/j.gastro.2023.06.032. Epub 2023 Jul 14. No abstract available. PMID 37453563
- [Result] Siegel EM, Ulrich CM, Poole EM, Holmes RS, Jacobsen PB, Shibata D. The effects of obesity and obesity-related conditions on colorectal cancer prognosis. Cancer Control. 2010 Jan;17(1):52-7. doi: 10.1177/107327481001700107. PMID 20010519
- [Result] Liu JJ, Druta M, Shibata D, Coppola D, Boler I, Elahi A, Reich RR, Siegel E, Extermann M. Metabolic syndrome and colorectal cancer: is hyperinsulinemia/insulin receptor-mediated angiogenesis a critical process? J Geriatr Oncol. 2014 Jan;5(1):40-8. doi: 10.1016/j.jgo.2013.11.004. Epub 2013 Dec 18. PMID 24484717
- [Result] Liesenfeld DB, Habermann N, Toth R, Owen RW, Frei E, Staffa J, Schrotz-King P, Klika KD, Ulrich CM. Changes in urinary metabolic profiles of colorectal cancer patients enrolled in a prospective cohort study (ColoCare). Metabolomics. 2015 Aug;11(4):998-1012. doi: 10.1007/s11306-014-0758-3. Epub 2014 Dec 20. PMID 29250455
- [Result] Karami S, Han Y, Pande M, Cheng I, Rudd J, Pierce BL, Nutter EL, Schumacher FR, Kote-Jarai Z, Lindstrom S, Witte JS, Fang S, Han J, Kraft P, Hunter DJ, Song F, Hung RJ, McKay J, Gruber SB, Chanock SJ, Risch A, Shen H, Haiman CA, Boardman L, Ulrich CM, Casey G, Peters U, Amin Al Olama A, Berchuck A, Berndt SI, Bezieau S, Brennan P, Brenner H, Brinton L, Caporaso N, Chan AT, Chang-Claude J, Christiani DC, Cunningham JM, Easton D, Eeles RA, Eisen T, Gala M, Gallinger SJ, Gayther SA, Goode EL, Gronberg H, Henderson BE, Houlston R, Joshi AD, Kury S, Landi MT, Le Marchand L, Muir K, Newcomb PA, Permuth-Wey J, Pharoah P, Phelan C, Potter JD, Ramus SJ, Risch H, Schildkraut J, Slattery ML, Song H, Wentzensen N, White E, Wiklund F, Zanke BW, Sellers TA, Zheng W, Chatterjee N, Amos CI, Doherty JA; GECCO and the GAME-ON Network: CORECT, DRIVE, ELLIPSE, FOCI, and TRICL. Telomere structure and maintenance gene variants and risk of five cancer types. Int J Cancer. 2016 Dec 15;139(12):2655-2670. doi: 10.1002/ijc.30288. Epub 2016 Sep 8. PMID 27459707
- [Result] Himbert C, Ose J, Delphan M, Ulrich CM. A systematic review of the interrelation between diet- and surgery-induced weight loss and vitamin D status. Nutr Res. 2017 Feb;38:13-26. doi: 10.1016/j.nutres.2016.12.004. Epub 2016 Dec 8. PMID 28381350
- [Result] Klett H, Balavarca Y, Toth R, Gigic B, Habermann N, Scherer D, Schrotz-King P, Ulrich A, Schirmacher P, Herpel E, Brenner H, Ulrich CM, Michels KB, Busch H, Boerries M. Robust prediction of gene regulation in colorectal cancer tissues from DNA methylation profiles. Epigenetics. 2018;13(4):386-397. doi: 10.1080/15592294.2018.1460034. Epub 2018 May 3. PMID 29697014
- [Result] Neumeyer S, Banbury BL, Arndt V, Berndt SI, Bezieau S, Bien SA, Buchanan DD, Butterbach K, Caan BJ, Campbell PT, Casey G, Chan AT, Chanock SJ, Dai JY, Gallinger S, Giovannucci EL, Giles GG, Grady WM, Hampe J, Hoffmeister M, Hopper JL, Hsu L, Jenkins MA, Joshi A, Larsson SC, Le Marchand L, Lindblom A, Moreno V, Lemire M, Li L, Lin Y, Offit K, Newcomb PA, Pharaoh PD, Potter JD, Qi L, Rennert G, Schafmayer C, Schoen RE, Slattery ML, Song M, Ulrich CM, Win AK, White E, Wolk A, Woods MO, Wu AH, Gruber SB, Brenner H, Peters U, Chang-Claude J. Mendelian randomisation study of age at menarche and age at menopause and the risk of colorectal cancer. Br J Cancer. 2018 Jun;118(12):1639-1647. doi: 10.1038/s41416-018-0108-8. Epub 2018 May 24. PMID 29795306
- [Result] Holowatyj AN, Ulrich CM, Lewis MA. Racial/Ethnic Patterns of Young-Onset Noncardia Gastric Cancer. Cancer Prev Res (Phila). 2019 Nov;12(11):771-780. doi: 10.1158/1940-6207.CAPR-19-0200. Epub 2019 Aug 16. PMID 31420363
- [Result] Hardikar S, Albrechtsen RD, Achaintre D, Lin T, Pauleck S, Playdon M, Holowatyj AN, Gigic B, Schrotz-King P, Boehm J, Habermann N, Brezina S, Gsur A, van Roekel EH, Weijenberg MP, Keski-Rahkonen P, Scalbert A, Ose J, Ulrich CM. Impact of Pre-blood Collection Factors on Plasma Metabolomic Profiles. Metabolites. 2020 May 21;10(5):213. doi: 10.3390/metabo10050213. PMID 32455751
- [Result] Geijsen AJMR, Ulvik A, Gigic B, Kok DE, van Duijnhoven FJB, Holowatyj AN, Brezina S, van Roekel EH, Baierl A, Bergmann MM, Bohm J, Bours MJL, Brenner H, Breukink SO, Bronner MP, Chang-Claude J, de Wilt JHW, Grady WM, Grunberger T, Gumpenberger T, Herpel E, Hoffmeister M, Huang LC, Jedrzkiewicz JD, Keulen ETP, Kiblawi R, Kolsch T, Koole JL, Kosma K, Kouwenhoven EA, Kruyt FM, Kvalheim G, Li CI, Lin T, Ose J, Pickron TB, Scaife CL, Schirmacher P, Schneider MA, Schrotz-King P, Singer MC, Swanson ER, van Duijvendijk P, van Halteren HK, van Zutphen M, Vickers K, Vogelaar FJ, Wesselink E, Habermann N, Ulrich AB, Ueland PM, Weijenberg MP, Gsur A, Ulrich CM, Kampman E. Circulating Folate and Folic Acid Concentrations: Associations With Colorectal Cancer Recurrence and Survival. JNCI Cancer Spectr. 2020 Jul 7;4(5):pkaa051. doi: 10.1093/jncics/pkaa051. eCollection 2020 Oct. PMID 33134831
- [Result] Tian Y, Kim AE, Bien SA, Lin Y, Qu C, Harrison TA, Carreras-Torres R, Diez-Obrero V, Dimou N, Drew DA, Hidaka A, Huyghe JR, Jordahl KM, Morrison J, Murphy N, Obon-Santacana M, Ulrich CM, Ose J, Peoples AR, Ruiz-Narvaez EA, Shcherbina A, Stern MC, Su YR, van Duijnhoven FJB, Arndt V, Baurley JW, Berndt SI, Bishop DT, Brenner H, Buchanan DD, Chan AT, Figueiredo JC, Gallinger S, Gruber SB, Harlid S, Hoffmeister M, Jenkins MA, Joshi AD, Keku TO, Larsson SC, Le Marchand L, Li L, Giles GG, Milne RL, Nan H, Nassir R, Ogino S, Budiarto A, Platz EA, Potter JD, Prentice RL, Rennert G, Sakoda LC, Schoen RE, Slattery ML, Thibodeau SN, Van Guelpen B, Visvanathan K, White E, Wolk A, Woods MO, Wu AH, Campbell PT, Casey G, Conti DV, Gunter MJ, Kundaje A, Lewinger JP, Moreno V, Newcomb PA, Pardamean B, Thomas DC, Tsilidis KK, Peters U, Gauderman WJ, Hsu L, Chang-Claude J. Genome-Wide Interaction Analysis of Genetic Variants With Menopausal Hormone Therapy for Colorectal Cancer Risk. J Natl Cancer Inst. 2022 Aug 8;114(8):1135-1148. doi: 10.1093/jnci/djac094. PMID 35512400
- [Result] Sleight AG, Crowder SL, Skarbinski J, Coen P, Parker NH, Hoogland AI, Gonzalez BD, Playdon MC, Cole S, Ose J, Murayama Y, Siegel EM, Figueiredo JC, Jim HSL. A New Approach to Understanding Cancer-Related Fatigue: Leveraging the 3P Model to Facilitate Risk Prediction and Clinical Care. Cancers (Basel). 2022 Apr 14;14(8):1982. doi: 10.3390/cancers14081982. PMID 35454890
- [Result] Shu X, Chen Z, Long J, Guo X, Yang Y, Qu C, Ahn YO, Cai Q, Casey G, Gruber SB, Huyghe JR, Jee SH, Jenkins MA, Jia WH, Jung KJ, Kamatani Y, Kim DH, Kim J, Kweon SS, Le Marchand L, Matsuda K, Matsuo K, Newcomb PA, Oh JH, Ose J, Oze I, Pai RK, Pan ZZ, Pharoah PDP, Playdon MC, Ren ZF, Schoen RE, Shin A, Shin MH, Shu XO, Sun X, Tangen CM, Tanikawa C, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Wolk A, Woods MO, Wu AH, Peters U, Zheng W. Large-scale Integrated Analysis of Genetics and Metabolomic Data Reveals Potential Links Between Lipids and Colorectal Cancer Risk. Cancer Epidemiol Biomarkers Prev. 2022 Jun 1;31(6):1216-1226. doi: 10.1158/1055-9965.EPI-21-1008. PMID 35266989
- [Result] Peoples AR, Oswald LB, Ose J, Daniels B, Himbert C, Hathaway CA, Gigic B, Kirchhoff AC, Lin T, Grossman D, Tward J, Varghese TK Jr, Figueiredo JC, Toriola AT, Beck A, Scaife C, Shibata D, LaStayo P, Gonzalez B, Salas K, Ashworth A, Matsen C, Christenson C, Ma DS, Colman H, Hunt JP, Jones KB, Lee CJ, Larson M, Onega T, Akerley WL, Li CI, Schneider M, Penedo FJ, Siegel EM, Tworoger SS, Ulrich CM. Impact of the COVID-19 pandemic on rural and urban cancer patients' experiences, health behaviors, and perceptions. J Rural Health. 2022 Sep;38(4):886-899. doi: 10.1111/jrh.12648. Epub 2022 Mar 3. PMID 35243690
- [Result] Pauleck S, Gigic B, Cawthon RM, Ose J, Peoples AR, Warby CA, Sinnott JA, Lin T, Boehm J, Schrotz-King P, Li CI, Shibata D, Siegel EM, Figueiredo JC, Toriola AT, Schneider M, Ulrich AB, Hoffmeister A, Ulrich CM, Hardikar S. Association of circulating leukocyte telomere length with survival in patients with colorectal cancer. J Geriatr Oncol. 2022 May;13(4):480-485. doi: 10.1016/j.jgo.2021.12.008. Epub 2022 Jan 5. PMID 34998722
- [Result] Jordahl KM, Shcherbina A, Kim AE, Su YR, Lin Y, Wang J, Qu C, Albanes D, Arndt V, Baurley JW, Berndt SI, Bien SA, Bishop DT, Bouras E, Brenner H, Buchanan DD, Budiarto A, Campbell PT, Carreras-Torres R, Casey G, Cenggoro TW, Chan AT, Conti DV, Dampier CH, Devall MA, Diez-Obrero V, Dimou N, Drew DA, Figueiredo JC, Gallinger S, Giles GG, Gruber SB, Gsur A, Gunter MJ, Hampel H, Harlid S, Harrison TA, Hidaka A, Hoffmeister M, Huyghe JR, Jenkins MA, Joshi AD, Keku TO, Larsson SC, Le Marchand L, Lewinger JP, Li L, Mahesworo B, Moreno V, Morrison JL, Murphy N, Nan H, Nassir R, Newcomb PA, Obon-Santacana M, Ogino S, Ose J, Pai RK, Palmer JR, Papadimitriou N, Pardamean B, Peoples AR, Pharoah PDP, Platz EA, Potter JD, Prentice RL, Rennert G, Ruiz-Narvaez E, Sakoda LC, Scacheri PC, Schmit SL, Schoen RE, Slattery ML, Stern MC, Tangen CM, Thibodeau SN, Thomas DC, Tian Y, Tsilidis KK, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Visvanathan K, Vodicka P, White E, Wolk A, Woods MO, Wu AH, Zemlianskaia N, Chang-Claude J, Gauderman WJ, Hsu L, Kundaje A, Peters U. Beyond GWAS of Colorectal Cancer: Evidence of Interaction with Alcohol Consumption and Putative Causal Variant for the 10q24.2 Region. Cancer Epidemiol Biomarkers Prev. 2022 May 4;31(5):1077-1089. doi: 10.1158/1055-9965.EPI-21-1003. PMID 35438744
- [Result] Holowatyj AN, Ose J, Gigic B, Lin T, Ulvik A, Geijsen AJMR, Brezina S, Kiblawi R, van Roekel EH, Baierl A, Bohm J, Bours MJL, Brenner H, Breukink SO, Chang-Claude J, de Wilt JHW, Grady WM, Grunberger T, Gumpenberger T, Herpel E, Hoffmeister M, Keulen ETP, Kok DE, Koole JL, Kosma K, Kouwenhoven EA, Kvalheim G, Li CI, Schirmacher P, Schrotz-King P, Singer MC, van Duijnhoven FJB, van Halteren HK, Vickers K, Vogelaar FJ, Warby CA, Wesselink E, Ueland PM, Ulrich AB, Schneider M, Habermann N, Kampman E, Weijenberg MP, Gsur A, Ulrich CM. Higher vitamin B6 status is associated with improved survival among patients with stage I-III colorectal cancer. Am J Clin Nutr. 2022 Aug 4;116(2):303-313. doi: 10.1093/ajcn/nqac090. PMID 35394006
- [Result] Hathaway CA, Bloomer AM, Oswald LB, Siegel EM, Peoples AR, Ulrich CM, Penedo FJ, Tworoger SS, Gonzalez BD. Factors associated with self-reported social isolation among patients with cancer during the COVID-19 pandemic. Health Psychol. 2022 Apr;41(4):311-318. doi: 10.1037/hea0001172. PMID 35324248
- [Result] Himbert C, Hathaway CA, Daniels B, Salas K, Ashworth A, Gigic B, Lin T, Viskochil R, Kirchhoff AC, Grossman D, Ose J, Tward J, Scaife C, Figueiredo JC, Toriola AT, Beck A, Shibata D, Gonzalez BD, Matsen C, Christenson C, Ma DS, Colman H, Hunt JP, Jones KB, Lee CJ, Larson M, Onega T, Akerley WL, Li CI, Schneider M, Penedo FJ, Siegel EM, Tworoger SS, Ulrich CM, Peoples AR. Factors associated with changes in exercise behaviors during the COVID-19 pandemic. Cancer Causes Control. 2022 Jul;33(7):939-950. doi: 10.1007/s10552-022-01580-z. Epub 2022 May 12. PMID 35554777
- [Result] Crowder SL, Playdon MC, Gudenkauf LM, Ose J, Gigic B, Greathouse L, Peoples AR, Sleight AG, Jim HSL, Figueiredo JC. A Molecular Approach to Understanding the Role of Diet in Cancer-Related Fatigue: Challenges and Future Opportunities. Nutrients. 2022 Apr 2;14(7):1496. doi: 10.3390/nu14071496. PMID 35406105
- [Result] Stewart KL, Gigic B, Himbert C, Warby CA, Ose J, Lin T, Schrotz-King P, Boehm J, Jordan KC, Metos J, Schneider M, Figueiredo JC, Li CI, Shibata D, Siegel E, Toriola AT, Hardikar S, Ulrich CM. Association of Sugar Intake with Inflammation- and Angiogenesis-Related Biomarkers in Newly Diagnosed Colorectal Cancer Patients. Nutr Cancer. 2022;74(5):1636-1643. doi: 10.1080/01635581.2021.1957133. Epub 2021 Aug 9. PMID 34369225
- [Result] Ose J, Gigic B, Hardikar S, Lin T, Himbert C, Warby CA, Peoples AR, Lindley CL, Boehm J, Schrotz-King P, Figueiredo JC, Toriola AT, Siegel EM, Li CI, Ulrich A, Schneider M, Shibata D, Ulrich CM. Presurgery Adhesion Molecules and Angiogenesis Biomarkers Are Differently Associated with Outcomes in Colon and Rectal Cancer: Results from the ColoCare Study. Cancer Epidemiol Biomarkers Prev. 2022 Aug 2;31(8):1650-1660. doi: 10.1158/1055-9965.EPI-22-0092. PMID 35667092
- [Result] Holthuijsen DDB, Bours MJL, Roekel EHV, Breukink SO, Janssen-Heijnen MLG, Keulen ETP, Ueland PM, Midttun O, Brezina S, Gigic B, Gsur A, Kok DE, Ose J, Ulrich CM, Weijenberg MP, Eussen SJPM. Longitudinal Associations of Adherence to the Dietary World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) and Dutch Healthy Diet (DHD) Recommendations with Plasma Kynurenines in Colorectal Cancer Survivors after Treatment. Nutrients. 2022 Dec 3;14(23):5151. doi: 10.3390/nu14235151. PMID 36501181
- [Result] Himbert C, Warby CA, Gigic B, Ose J, Lin T, Viskochil R, Peoples AR, Ashworth A, Schrotz-King P, Scaife CL, Cohan JN, Jedrzkiewicz J, Schirmacher P, Grady WM, Cohen SA, Krane M, Figueiredo JC, Toriola AT, Siegel EM, Shibata D, Round JL, Huang LC, Li CI, Schneider M, Ulrich A, Hardikar S, Ulrich CM. Associations of Individual and Combined Physical Activity and Body Mass Index Groups with Proinflammatory Biomarkers among Colorectal Cancer Patients. Cancer Epidemiol Biomarkers Prev. 2022 Dec 5;31(12):2148-2156. doi: 10.1158/1055-9965.EPI-22-0681. PMID 36099423
- [Result] Himbert C, Stephens WZ, Gigic B, Hardikar S, Holowatyj AN, Lin T, Ose J, Swanson E, Ashworth A, Warby CA, Peoples AR, Nix D, Jedrzkiewicz J, Bronner M, Pickron B, Scaife C, Cohan JN, Schrotz-King P, Habermann N, Boehm J, Hullar M, Figueiredo JC, Toriola AT, Siegel EM, Li CI, Ulrich AB, Shibata D, Boucher K, Huang LC, Schneider M, Round JL, Ulrich CM. Differences in the gut microbiome by physical activity and BMI among colorectal cancer patients. Am J Cancer Res. 2022 Oct 15;12(10):4789-4801. eCollection 2022. PMID 36381318
- [Result] Gigic B, van Roekel E, Holowatyj AN, Brezina S, Geijsen AJMR, Ulvik A, Ose J, Koole JL, Damerell V, Kiblawi R, Gumpenberger T, Lin T, Kvalheim G, Koelsch T, Kok DE, van Duijnhoven FJ, Bours MJ, Baierl A, Li CI, Grady W, Vickers K, Habermann N, Schneider M, Kampman E, Ueland PM, Ulrich A, Weijenberg M, Gsur A, Ulrich C; FOCUS Consortium. Cohort profile: Biomarkers related to folate-dependent one-carbon metabolism in colorectal cancer recurrence and survival - the FOCUS Consortium. BMJ Open. 2022 Dec 22;12(12):e062930. doi: 10.1136/bmjopen-2022-062930. PMID 36549742
- [Result] Luo Y, Tsuchiya KD, Il Park D, Fausel R, Kanngurn S, Welcsh P, Dzieciatkowski S, Wang J, Grady WM. RET is a potential tumor suppressor gene in colorectal cancer. Oncogene. 2013 Apr 18;32(16):2037-47. doi: 10.1038/onc.2012.225. Epub 2012 Jul 2. PMID 22751117
- [Result] Lao VV, Welcsh P, Luo Y, Carter KT, Dzieciatkowski S, Dintzis S, Meza J, Sarvetnick NE, Monnat RJ Jr, Loeb LA, Grady WM. Altered RECQ Helicase Expression in Sporadic Primary Colorectal Cancers. Transl Oncol. 2013 Aug 1;6(4):458-69. doi: 10.1593/tlo.13238. Print 2013 Aug. PMID 23908689
- [Result] Luo Y, Kaz AM, Kanngurn S, Welsch P, Morris SM, Wang J, Lutterbaugh JD, Markowitz SD, Grady WM. NTRK3 is a potential tumor suppressor gene commonly inactivated by epigenetic mechanisms in colorectal cancer. PLoS Genet. 2013;9(7):e1003552. doi: 10.1371/journal.pgen.1003552. Epub 2013 Jul 11. PMID 23874207
- [Result] Yu M, Carter KT, Makar KW, Vickers K, Ulrich CM, Schoen RE, Brenner D, Markowitz SD, Grady WM. MethyLight droplet digital PCR for detection and absolute quantification of infrequently methylated alleles. Epigenetics. 2015;10(9):803-9. doi: 10.1080/15592294.2015.1068490. Epub 2015 Jul 17. PMID 26186366
- [Result] Toth R, Scherer D, Kelemen LE, Risch A, Hazra A, Balavarca Y, Issa JJ, Moreno V, Eeles RA, Ogino S, Wu X, Ye Y, Hung RJ, Goode EL, Ulrich CM; OCAC, CORECT, TRICL, ELLIPSE, DRIVE, and GAME-ON consortia. Genetic Variants in Epigenetic Pathways and Risks of Multiple Cancers in the GAME-ON Consortium. Cancer Epidemiol Biomarkers Prev. 2017 Jun;26(6):816-825. doi: 10.1158/1055-9965.EPI-16-0728. Epub 2017 Jan 23. PMID 28115406
- [Result] Dimitrakopoulou VI, Tsilidis KK, Haycock PC, Dimou NL, Al-Dabhani K, Martin RM, Lewis SJ, Gunter MJ, Mondul A, Shui IM, Theodoratou E, Nimptsch K, Lindstrom S, Albanes D, Kuhn T, Key TJ, Travis RC, Vimaleswaran KS; GECCO Consortium; PRACTICAL Consortium; GAME-ON Network (CORECT, DRIVE, ELLIPSE, FOCI-OCAC, TRICL-ILCCO); Kraft P, Pierce BL, Schildkraut JM. Circulating vitamin D concentration and risk of seven cancers: Mendelian randomisation study. BMJ. 2017 Oct 31;359:j4761. doi: 10.1136/bmj.j4761. PMID 29089348
- [Result] Matas J, Kohrn B, Fredrickson J, Carter K, Yu M, Wang T, Gui X, Soussi T, Moreno V, Grady WM, Peinado MA, Risques RA. Colorectal Cancer Is Associated with the Presence of Cancer Driver Mutations in Normal Colon. Cancer Res. 2022 Apr 15;82(8):1492-1502. doi: 10.1158/0008-5472.CAN-21-3607. PMID 35425963
- [Result] Ose DJ, Viskochil R, Holowatyj AN, Larson M, Wilson D, Dunson WA, Deshmukh VG, Butcher JR, Taylor BR, Svoboda K, Leiser J, Tingey B, Haaland B, Wetter DW, Fisher SJ, Hashibe M, Ulrich CM. Understanding the Prevalence of Prediabetes and Diabetes in Patients With Cancer in Clinical Practice: A Real-World Cohort Study. J Natl Compr Canc Netw. 2021 Mar 10;19(6):709-718. doi: 10.6004/jnccn.2020.7653. PMID 34129522
- [Result] Holowatyj AN, Gigic B, Warby CA, Ose J, Lin T, Schrotz-King P, Ulrich CM, Bernard JJ. The Use of Human Serum Samples to Study Malignant Transformation: A Pilot Study. Cells. 2021 Oct 6;10(10):2670. doi: 10.3390/cells10102670. PMID 34685650
- [Result] Holowatyj AN, Viskochil R, Ose D, Tingey B, Haaland B, Wilson D, Larson M, Feltz S, Lewis MA, Colman H, Ulrich CM. Diabetes, Body Fatness, and Insulin Prescription Among Adolescents and Young Adults with Cancer. J Adolesc Young Adult Oncol. 2021 Apr;10(2):217-225. doi: 10.1089/jayao.2020.0071. Epub 2020 Jul 29. PMID 32749900
- [Result] Grady WM, Yu M, Markowitz SD. Epigenetic Alterations in the Gastrointestinal Tract: Current and Emerging Use for Biomarkers of Cancer. Gastroenterology. 2021 Feb;160(3):690-709. doi: 10.1053/j.gastro.2020.09.058. Epub 2020 Dec 3. PMID 33279516
- [Result] Nounu A, Richmond RC, Stewart ID, Surendran P, Wareham NJ, Butterworth A, Weinstein SJ, Albanes D, Baron JA, Hopper JL, Figueiredo JC, Newcomb PA, Lindor NM, Casey G, Platz EA, Marchand LL, Ulrich CM, Li CI, van Dujinhoven FJB, Gsur A, Campbell PT, Moreno V, Vodicka P, Vodickova L, Amitay E, Alwers E, Chang-Claude J, Sakoda LC, Slattery ML, Schoen RE, Gunter MJ, Castellvi-Bel S, Kim HR, Kweon SS, Chan AT, Li L, Zheng W, Bishop DT, Buchanan DD, Giles GG, Gruber SB, Rennert G, Stadler ZK, Harrison TA, Lin Y, Keku TO, Woods MO, Schafmayer C, Van Guelpen B, Gallinger S, Hampel H, Berndt SI, Pharoah PDP, Lindblom A, Wolk A, Wu AH, White E, Peters U, Drew DA, Scherer D, Bermejo JL, Brenner H, Hoffmeister M, Williams AC, Relton CL. Salicylic Acid and Risk of Colorectal Cancer: A Two-Sample Mendelian Randomization Study. Nutrients. 2021 Nov 21;13(11):4164. doi: 10.3390/nu13114164. PMID 34836419
- [Result] Dimou N, Yarmolinsky J, Bouras E, Tsilidis KK, Martin RM, Lewis SJ, Gram IT, Bakker MF, Brenner H, Figueiredo JC, Fortner RT, Gruber SB, van Guelpen B, Hsu L, Kaaks R, Kweon SS, Lin Y, Lindor NM, Newcomb PA, Sanchez MJ, Severi G, Tindle HA, Tumino R, Weiderpass E, Gunter MJ, Murphy N. Causal Effects of Lifetime Smoking on Breast and Colorectal Cancer Risk: Mendelian Randomization Study. Cancer Epidemiol Biomarkers Prev. 2021 May;30(5):953-964. doi: 10.1158/1055-9965.EPI-20-1218. Epub 2021 Mar 2. PMID 33653810
- [Result] Himbert C, Figueiredo JC, Shibata D, Ose J, Lin T, Huang LC, Peoples AR, Scaife CL, Pickron B, Lambert L, Cohan JN, Bronner M, Felder S, Sanchez J, Dessureault S, Coppola D, Hoffman DM, Nasseri YF, Decker RW, Zaghiyan K, Murrell ZA, Hendifar A, Gong J, Firoozmand E, Gangi A, Moore BA, Cologne KG, El-Masry MS, Hinkle N, Monroe J, Mutch M, Bernadt C, Chatterjee D, Sinanan M, Cohen SA, Wallin U, Grady WM, Lampe PD, Reddi D, Krane M, Fichera A, Moonka R, Herpel E, Schirmacher P, Kloor M, von Knebel-Doeberitz M, Nattenmueller J, Kauczor HU, Swanson E, Jedrzkiewicz J, Schmit SL, Gigic B, Ulrich AB, Toriola AT, Siegel EM, Li CI, Ulrich CM, Hardikar S. Clinical Characteristics and Outcomes of Colorectal Cancer in the ColoCare Study: Differences by Age of Onset. Cancers (Basel). 2021 Jul 29;13(15):3817. doi: 10.3390/cancers13153817. PMID 34359718
- [Result] Lu Y, Kweon SS, Cai Q, Tanikawa C, Shu XO, Jia WH, Xiang YB, Huyghe JR, Harrison TA, Kim J, Shin A, Kim DH, Matsuo K, Jee SH, Guo X, Wen W, Shi J, Li B, Wang N, Shin MH, Li HL, Ren Z, Oh JH, Oze I, Ahn YO, Jung KJ, Gao J, Gao YT, Pan ZZ, Kamatani Y, Chan AT, Gsur A, Hampe J, Le Marchand L, Li L, Lindblom A, Moreno V, Newcomb PA, Offit K, Pharoah PDP, van Duijnhoven FJB, Van Guelpen B, Vodicka P, Weinstein SJ, Wolk A, Wu AH, Hsu L, Zeng YX, Long J, Peters U, Matsuda K, Zheng W. Identification of Novel Loci and New Risk Variant in Known Loci for Colorectal Cancer Risk in East Asians. Cancer Epidemiol Biomarkers Prev. 2020 Feb;29(2):477-486. doi: 10.1158/1055-9965.EPI-19-0755. Epub 2019 Dec 11. PMID 31826910
- [Result] Murphy N, Carreras-Torres R, Song M, Chan AT, Martin RM, Papadimitriou N, Dimou N, Tsilidis KK, Banbury B, Bradbury KE, Besevic J, Rinaldi S, Riboli E, Cross AJ, Travis RC, Agnoli C, Albanes D, Berndt SI, Bezieau S, Bishop DT, Brenner H, Buchanan DD, Onland-Moret NC, Burnett-Hartman A, Campbell PT, Casey G, Castellvi-Bel S, Chang-Claude J, Chirlaque MD, de la Chapelle A, English D, Figueiredo JC, Gallinger SJ, Giles GG, Gruber SB, Gsur A, Hampe J, Hampel H, Harrison TA, Hoffmeister M, Hsu L, Huang WY, Huyghe JR, Jenkins MA, Keku TO, Kuhn T, Kweon SS, Le Marchand L, Li CI, Li L, Lindblom A, Martin V, Milne RL, Moreno V, Newcomb PA, Offit K, Ogino S, Ose J, Perduca V, Phipps AI, Platz EA, Potter JD, Qu C, Rennert G, Sakoda LC, Schafmayer C, Schoen RE, Slattery ML, Tangen CM, Ulrich CM, van Duijnhoven FJB, Van Guelpen B, Visvanathan K, Vodicka P, Vodickova L, Vymetalkova V, Wang H, White E, Wolk A, Woods MO, Wu AH, Zheng W, Peters U, Gunter MJ. Circulating Levels of Insulin-like Growth Factor 1 and Insulin-like Growth Factor Binding Protein 3 Associate With Risk of Colorectal Cancer Based on Serologic and Mendelian Randomization Analyses. Gastroenterology. 2020 Apr;158(5):1300-1312.e20. doi: 10.1053/j.gastro.2019.12.020. Epub 2019 Dec 27. PMID 31884074
- [Result] Scherer D, Deutelmoser H, Balavarca Y, Toth R, Habermann N, Buck K, Kap EJ, Botma A, Seibold P, Jansen L, Lorenzo Bermejo J, Weigl K, Benner A, Hoffmeister M, Ulrich A, Brenner H, Burwinkel B, Chang-Claude J, Ulrich CM. Polymorphisms in the Angiogenesis-Related Genes EFNB2, MMP2 and JAG1 Are Associated with Survival of Colorectal Cancer Patients. Int J Mol Sci. 2020 Jul 29;21(15):5395. doi: 10.3390/ijms21155395. PMID 32751332
- [Result] Khankari NK, Banbury BL, Borges MC, Haycock P, Albanes D, Arndt V, Berndt SI, Bezieau S, Brenner H, Campbell PT, Casey G, Chan AT, Chang-Claude J, Conti DV, Cotterchio M, English DR, Figueiredo JC, Giles GG, Giovannucci EL, Gunter MJ, Hampe J, Hoffmeister M, Hopper JL, Jenkins MA, Joshi AD, Marchand LL, Lemire M, Li CI, Li L, Lindblom A, Martin V, Moreno V, Newcomb PA, Offit K, Pharoah PDP, Rennert G, Sakoda LC, Schafmayer C, Schmit SL, Slattery ML, Song M, Thibodeau SN, Ulrich CM, Weinstein SJ, White E, Win AK, Wolk A, Woods MO, Wu AH, Cai Q, Denny JC, Edwards TL, Murff HJ, Gruber SB, Peters U, Zheng W. Mendelian Randomization of Circulating Polyunsaturated Fatty Acids and Colorectal Cancer Risk. Cancer Epidemiol Biomarkers Prev. 2020 Apr;29(4):860-870. doi: 10.1158/1055-9965.EPI-19-0891. Epub 2020 Feb 12. PMID 32051193
- [Result] Himbert C, Klossner N, Coletta AM, Barnes CA, Wiskemann J, LaStayo PC, Varghese TK Jr, Ulrich CM. Exercise and lung cancer surgery: A systematic review of randomized-controlled trials. Crit Rev Oncol Hematol. 2020 Dec;156:103086. doi: 10.1016/j.critrevonc.2020.103086. Epub 2020 Sep 13. PMID 33038630
- [Result] Jiang Y, Spurny M, Schubel R, Nonnenmacher T, Schlett CL, von Stackelberg O, Ulrich CM, Kaaks R, Kauczor HU, Kuhn T, Nattenmuller J. Changes in Pancreatic Fat Content Following Diet-Induced Weight Loss. Nutrients. 2019 Apr 23;11(4):912. doi: 10.3390/nu11040912. PMID 31018616
- [Result] Geijsen AJMR, Brezina S, Keski-Rahkonen P, Baierl A, Bachleitner-Hofmann T, Bergmann MM, Boehm J, Brenner H, Chang-Claude J, van Duijnhoven FJB, Gigic B, Gumpenberger T, Hofer P, Hoffmeister M, Holowatyj AN, Karner-Hanusch J, Kok DE, Leeb G, Ulvik A, Robinot N, Ose J, Stift A, Schrotz-King P, Ulrich AB, Ueland PM, Kampman E, Scalbert A, Habermann N, Gsur A, Ulrich CM. Plasma metabolites associated with colorectal cancer: A discovery-replication strategy. Int J Cancer. 2019 Sep 1;145(5):1221-1231. doi: 10.1002/ijc.32146. Epub 2019 Feb 14. PMID 30665271
- [Result] Guo Y, Ayers JL, Carter KT, Wang T, Maden SK, Edmond D, Newcomb P P, Li C, Ulrich C, Yu M, Grady WM. Senescence-associated tissue microenvironment promotes colon cancer formation through the secretory factor GDF15. Aging Cell. 2019 Dec;18(6):e13013. doi: 10.1111/acel.13013. Epub 2019 Aug 6. PMID 31389184
- [Result] Sheth H, Northwood E, Ulrich CM, Scherer D, Elliott F, Barrett JH, Forman D, Wolf CR, Smith G, Jackson MS, Santibanez-Koref M, Haile R, Casey G, Jenkins M, Win AK, Hopper JL, Marchand LL, Lindor NM, Thibodeau SN, Potter JD, Burn J, Bishop DT. Interaction between polymorphisms in aspirin metabolic pathways, regular aspirin use and colorectal cancer risk: A case-control study in unselected white European populations. PLoS One. 2018 Feb 9;13(2):e0192223. doi: 10.1371/journal.pone.0192223. eCollection 2018. PMID 29425227
- [Result] Ulrich CM, Himbert C, Boucher K, Wetter DW, Hess R, Kim J, Lundberg K, Ligibel JA, Barnes CA, Rushton B, Marcus R, Finlayson SRG, LaStayo PC, Varghese TK. Precision-Exercise-Prescription in patients with lung cancer undergoing surgery: rationale and design of the PEP study trial. BMJ Open. 2018 Dec 16;8(12):e024672. doi: 10.1136/bmjopen-2018-024672. PMID 30559162
- [Result] Lauby-Secretan B, Scoccianti C, Loomis D, Grosse Y, Bianchini F, Straif K; International Agency for Research on Cancer Handbook Working Group. Body Fatness and Cancer--Viewpoint of the IARC Working Group. N Engl J Med. 2016 Aug 25;375(8):794-8. doi: 10.1056/NEJMsr1606602. No abstract available. PMID 27557308
- [Result] Peruchet-Noray L, Sedlmeier AM, Dimou N, Baurecht H, Fervers B, Fontvieille E, Konzok J, Tsilidis KK, Christakoudi S, Jansana A, Cordova R, Bohmann P, Stein MJ, Weber A, Bezieau S, Brenner H, Chan AT, Cheng I, Figueiredo JC, Garcia-Etxebarria K, Moreno V, Newton CC, Schmit SL, Song M, Ulrich CM, Ferrari P, Viallon V, Carreras-Torres R, Gunter MJ, Freisling H. Tissue-specific genetic variation suggests distinct molecular pathways between body shape phenotypes and colorectal cancer. Sci Adv. 2024 Apr 19;10(16):eadj1987. doi: 10.1126/sciadv.adj1987. Epub 2024 Apr 19. PMID 38640244
- [Result] Chen Z, Guo X, Tao R, Huyghe JR, Law PJ, Fernandez-Rozadilla C, Ping J, Jia G, Long J, Li C, Shen Q, Xie Y, Timofeeva MN, Thomas M, Schmit SL, Diez-Obrero V, Devall M, Moratalla-Navarro F, Fernandez-Tajes J, Palles C, Sherwood K, Briggs SEW, Svinti V, Donnelly K, Farrington SM, Blackmur J, Vaughan-Shaw PG, Shu XO, Lu Y, Broderick P, Studd J, Harrison TA, Conti DV, Schumacher FR, Melas M, Rennert G, Obon-Santacana M, Martin-Sanchez V, Oh JH, Kim J, Jee SH, Jung KJ, Kweon SS, Shin MH, Shin A, Ahn YO, Kim DH, Oze I, Wen W, Matsuo K, Matsuda K, Tanikawa C, Ren Z, Gao YT, Jia WH, Hopper JL, Jenkins MA, Win AK, Pai RK, Figueiredo JC, Haile RW, Gallinger S, Woods MO, Newcomb PA, Duggan D, Cheadle JP, Kaplan R, Kerr R, Kerr D, Kirac I, Bohm J, Mecklin JP, Jousilahti P, Knekt P, Aaltonen LA, Rissanen H, Pukkala E, Eriksson JG, Cajuso T, Hanninen U, Kondelin J, Palin K, Tanskanen T, Renkonen-Sinisalo L, Mannisto S, Albanes D, Weinstein SJ, Ruiz-Narvaez E, Palmer JR, Buchanan DD, Platz EA, Visvanathan K, Ulrich CM, Siegel E, Brezina S, Gsur A, Campbell PT, Chang-Claude J, Hoffmeister M, Brenner H, Slattery ML, Potter JD, Tsilidis KK, Schulze MB, Gunter MJ, Murphy N, Castells A, Castellvi-Bel S, Moreira L, Arndt V, Shcherbina A, Bishop DT, Giles GG, Southey MC, Idos GE, McDonnell KJ, Abu-Ful Z, Greenson JK, Shulman K, Lejbkowicz F, Offit K, Su YR, Steinfelder R, Keku TO, van Guelpen B, Hudson TJ, Hampel H, Pearlman R, Berndt SI, Hayes RB, Martinez ME, Thomas SS, Pharoah PDP, Larsson SC, Yen Y, Lenz HJ, White E, Li L, Doheny KF, Pugh E, Shelford T, Chan AT, Cruz-Correa M, Lindblom A, Hunter DJ, Joshi AD, Schafmayer C, Scacheri PC, Kundaje A, Schoen RE, Hampe J, Stadler ZK, Vodicka P, Vodickova L, Vymetalkova V, Edlund CK, Gauderman WJ, Shibata D, Toland A, Markowitz S, Kim A, Chanock SJ, van Duijnhoven F, Feskens EJM, Sakoda LC, Gago-Dominguez M, Wolk A, Pardini B, FitzGerald LM, Lee SC, Ogino S, Bien SA, Kooperberg C, Li CI, Lin Y, Prentice R, Qu C, Bezieau S, Yamaji T, Sawada N, Iwasaki M, Le Marchand L, Wu AH, Qu C, McNeil CE, Coetzee G, Hayward C, Deary IJ, Harris SE, Theodoratou E, Reid S, Walker M, Ooi LY, Lau KS, Zhao H, Hsu L, Cai Q, Dunlop MG, Gruber SB, Houlston RS, Moreno V, Casey G, Peters U, Tomlinson I, Zheng W. Fine-mapping analysis including over 254,000 East Asian and European descendants identifies 136 putative colorectal cancer susceptibility genes. Nat Commun. 2024 Apr 26;15(1):3557. doi: 10.1038/s41467-024-47399-x. PMID 38670944
- [Result] Wang C, Ma A, Li Y, McNutt ME, Zhang S, Zhu J, Hoyd R, Wheeler CE, Robinson LA, Chan CHF, Zakharia Y, Dodd RD, Ulrich CM, Hardikar S, Churchman ML, Tarhini AA, Singer EA, Ikeguchi AP, McCarter MD, Denko N, Tinoco G, Husain M, Jin N, Osman AEG, Eljilany I, Tan AC, Coleman SS, Denko L, Riedlinger G, Schneider BP, Spakowicz D, Ma Q; exORIEN Consortium. A Bioinformatics Tool for Identifying Intratumoral Microbes from the ORIEN Dataset. Cancer Res Commun. 2024 Feb 5;4(2):293-302. doi: 10.1158/2767-9764.CRC-23-0213. PMID 38259095
- [Result] Papadimitriou N, Kim A, Kawaguchi ES, Morrison J, Diez-Obrero V, Albanes D, Berndt SI, Bezieau S, Bien SA, Bishop DT, Bouras E, Brenner H, Buchanan DD, Campbell PT, Carreras-Torres R, Chan AT, Chang-Claude J, Conti DV, Devall MA, Dimou N, Drew DA, Gruber SB, Harrison TA, Hoffmeister M, Huyghe JR, Joshi AD, Keku TO, Kundaje A, Kury S, Le Marchand L, Lewinger JP, Li L, Lynch BM, Moreno V, Newton CC, Obon-Santacana M, Ose J, Pellatt AJ, Peoples AR, Platz EA, Qu C, Rennert G, Ruiz-Narvaez E, Shcherbina A, Stern MC, Su YR, Thomas DC, Thomas CE, Tian Y, Tsilidis KK, Ulrich CM, Um CY, Visvanathan K, Wang J, White E, Woods MO, Schmit SL, Macrae F, Potter JD, Hopper JL, Peters U, Murphy N, Hsu L, Gunter MJ, Gauderman WJ. Genome-wide interaction study of dietary intake of fibre, fruits, and vegetables with risk of colorectal cancer. EBioMedicine. 2024 Jun;104:105146. doi: 10.1016/j.ebiom.2024.105146. Epub 2024 May 14. PMID 38749303
- [Result] Oswald LB, Bloomer A, Li X, Jean-Baptiste E, Trujillo G, Felder S, Small BJ, Ose J, Hardikar S, Strehli I, Huang LC, Mooney K, Mutch MG, Chao D, Cohen SA, Karchi M, Wood EH, Damerell V, Lorona NC, Gong J, Toriola AT, Li CI, Shibata D, Schneider M, Gigic B, Figueiredo JC, Jim HSL, Ulrich CM, Siegel EM. Functional quality of life among newly diagnosed young adult colorectal cancer survivors compared to older adults: results from the ColoCare Study. Support Care Cancer. 2024 Apr 19;32(5):298. doi: 10.1007/s00520-024-08511-5. PMID 38639810
- [Result] Assmann ES, Ose J, Hathaway CA, Oswald LB, Hardikar S, Himbert C, Chellam V, Lin T, Daniels B, Kirchhoff AC, Gigic B, Grossman D, Tward J, Varghese TK Jr, Shibata D, Figueiredo JC, Toriola AT, Beck A, Scaife C, Barnes CA, Matsen C, Ma DS, Colman H, Hunt JP, Jones KB, Lee CJ, Larson M, Onega T, Akerley WL, Li CI, Grady WM, Schneider M, Dinkel A, Islam JY, Gonzalez BD, Otto AK, Penedo FJ, Siegel EM, Tworoger SS, Ulrich CM, Peoples AR. Risk factors and health behaviors associated with loneliness among cancer survivors during the COVID-19 pandemic. J Behav Med. 2024 Jun;47(3):405-421. doi: 10.1007/s10865-023-00465-z. Epub 2024 Feb 28. PMID 38418709
- [Result] Otto AK, Prinsloo S, Natori A, Wagner RW, Gomez TI, Ochoa JM, Tworoger SS, Ulrich CM, Ahmed S, McQuade JL, Peoples AR, Antoni MH, Bower JE, Cohen L, Penedo FJ. Impact of COVID-19-related experiences on health-related quality of life in cancer survivors in the United States. PLoS One. 2024 Mar 14;19(3):e0297077. doi: 10.1371/journal.pone.0297077. eCollection 2024. PMID 38484002
- [Result] Wagner RW, Natori A, Prinsloo S, Otto AK, Saez-Clarke E, Ochoa JM, Tworoger SS, Ulrich CM, Hathaway CA, Ahmed S, McQuade JL, Peoples AR, Antoni MH, Penedo FJ, Cohen L. The role of area deprivation index in health care disruptions among cancer survivors during the SARS-CoV-2 pandemic. Public Health. 2024 Jul;232:52-60. doi: 10.1016/j.puhe.2024.04.007. Epub 2024 May 11. PMID 38735226
- [Result] Holthuijsen DDB, van Roekel EH, Bours MJL, Ueland PM, Breukink SO, Janssen-Heijnen MLG, Keulen ETP, Gigic B, Gsur A, Meyer K, Ose J, Ulvik A, Weijenberg MP, Eussen SJPM. Longitudinal associations of plasma kynurenines and ratios with anxiety and depression scores in colorectal cancer survivors up to 12 months post-treatment. Psychoneuroendocrinology. 2024 May;163:106981. doi: 10.1016/j.psyneuen.2024.106981. Epub 2024 Jan 26. PMID 38335827
- [Result] Holthuijsen DDB, van Roekel EH, Bours MJL, Ueland PM, Breukink SO, Janssen-Heijnen MLG, Keulen ETP, Brezina S, Gigic B, Peoples AR, Ulrich CM, Ulvik A, Weijenberg MP, Eussen SJPM. Longitudinal associations of plasma kynurenines and ratios with fatigue and quality of life in colorectal cancer survivors up to 12 months post-treatment. Int J Cancer. 2024 Oct 1;155(7):1172-1190. doi: 10.1002/ijc.34992. Epub 2024 May 23. PMID 38783597
- [Result] Benej M, Hoyd R, Kreamer M, Wheeler CE, Grencewicz DJ, Choueiry F, Chan CHF, Zakharia Y, Ma Q, Dodd RD, Ulrich CM, Hardikar S, Churchman ML, Tarhini AA, Robinson LA, Singer EA, Ikeguchi AP, McCarter MD, Tinoco G, Husain M, Jin N, Tan AC, Osman AEG, Eljilany I, Riedlinger G, Schneider BP, Benejova K, Kery M, Papandreou I, Zhu J, Denko N, Spakowicz D; exORIEN Consortium. The Tumor Microbiome Reacts to Hypoxia and Can Influence Response to Radiation Treatment in Colorectal Cancer. Cancer Res Commun. 2024 Jul 1;4(7):1690-1701. doi: 10.1158/2767-9764.CRC-23-0367. PMID 38904265
- [Result] Drew DA, Kim AE, Lin Y, Qu C, Morrison J, Lewinger JP, Kawaguchi E, Wang J, Fu Y, Zemlianskaia N, Diez-Obrero V, Bien SA, Dimou N, Albanes D, Baurley JW, Wu AH, Buchanan DD, Potter JD, Prentice RL, Harlid S, Arndt V, Barry EL, Berndt SI, Bouras E, Brenner H, Budiarto A, Burnett-Hartman A, Campbell PT, Carreras-Torres R, Casey G, Chang-Claude J, Conti DV, Devall MAM, Figueiredo JC, Gruber SB, Gsur A, Gunter MJ, Harrison TA, Hidaka A, Hoffmeister M, Huyghe JR, Jenkins MA, Jordahl KM, Kundaje A, Le Marchand L, Li L, Lynch BM, Murphy N, Nassir R, Newcomb PA, Newton CC, Obon-Santacana M, Ogino S, Ose J, Pai RK, Palmer JR, Papadimitriou N, Pardamean B, Pellatt AJ, Peoples AR, Platz EA, Rennert G, Ruiz-Narvaez E, Sakoda LC, Scacheri PC, Schmit SL, Schoen RE, Stern MC, Su YR, Thomas DC, Tian Y, Tsilidis KK, Ulrich CM, Um CY, van Duijnhoven FJB, Van Guelpen B, White E, Hsu L, Moreno V, Peters U, Chan AT, Gauderman WJ. Two genome-wide interaction loci modify the association of nonsteroidal anti-inflammatory drugs with colorectal cancer. Sci Adv. 2024 May 31;10(22):eadk3121. doi: 10.1126/sciadv.adk3121. Epub 2024 May 29. PMID 38809988
- [Derived] Peoples AR, Damerell V, Ose J, Siegel EM, Lin T, Hardikar S, Himbert C, Ilozumba MN, Schrotz-King P, Crowder SL, Toriola AT, Shibata D, Li CI, Byrd DA, Assmann ES, Jim HSL, Figueiredo JC, Ulrich CM, Gigic B. Association of Sleep Disturbance With Survival After Colorectal Cancer Diagnosis: Results From the ColoCare Study. Cancer Med. 2026 Feb;15(2):e71576. doi: 10.1002/cam4.71576. PMID 41588841
- [Derived] Hausmann O, Schobert PP, Ose J, Himbert C, Pletneva M, Jedrzkiewicz J, Nguyen A, Lin T, Warby CA, Hardikar S, Peoples AR, Strehli I, Huang LC, Cohan JN, Pickron B, Scaife C, Li CI, Grady WM, Shibata D, Toriola AT, Schneider M, Figueiredo JC, Siegel EM, Gigic B, Herzig S, Ilozumba MN, Ulrich CM. Associations of Biomarkers of Systemic Inflammation, Angiogenesis, and Cell-to-Cell Adhesion With Tumor Budding Among Early-Onset and Later-Onset Colorectal Cancer Patients. Cancer Med. 2025 Sep;14(18):e71267. doi: 10.1002/cam4.71267. PMID 40985344